## **Statistical Analysis Plan**

### **GLORIA**

The Glucocorticoid Low-dose Outcome in RheumatoId Arthritis Study

Comparing the cost-effectiveness and safety of additional low-dose glucocorticoid in treatment strategies for elderly patients with rheumatoid arthritis

Sponsor: VU University Medical Center

De Boelelaan 1117 1081 HV Amsterdam The Netherlands

Author: VU University Medical Center

Department of Epidemiology and Biostatistics &

Amsterdam Rheumatology and immunology Center, location VU University Medical

Center

Amsterdam, Netherlands

Date: March 2, 2021

Version: 1.0

## Sign-off signatures

| Author: | Linda Hartman | | | |
|---|---|---|---|---|
| | PhD student | | | |
| | | Signature | C | ate |
| Peer review: | Leonie Middelink | | | |
| | Project Operational Lead | | | |
| | | Signature | Г | )ate |
| | | Signature | _ | Juic |
| Approved by: | Maarten Boers | | | |
| | Project leader and Principal Investigat | or | | |
| | 1. / | | 02 Mar 2021 | |
| | Lu. L | Signature | 02-Mar-2021 | ate |
| Approved by: | | | | |
| прргочей бу. | Statistician | | | |
| | | Signaturo | Γ | ) ata |
| | | Jigilatule | L | ouc. |

#### **Table of contents**

| L | ist of a | bbrev | viations and definitions | 5 |
|---|---|---|---|---|
| 1 | Intro | ducti | ion | 6 |
| | 1.1 | Stuc | ly population | 6 |
| | 1.2 | Stuc | ly design | 6 |
| | 1.3 | Prim | nary and secondary study objectives | 8 |
| | 1.3. | .1 | Primary objectives | 8 |
| | 1.3. | .2 | Secondary objectives | 8 |
| | 1.4 | Prim | nary and secondary endpoints | 8 |
| | 1.4. | .1 | Primary endpoints | 8 |
| | 1.4. | .2 | Secondary endpoints | 10 |
| 2 | Anal | vsis p | opulations | 12 |
| _ | 2.1 | | nt-to-treat population | |
| | 2.2 | | protocol population, also excluding initial changes in antirheumatic medication | |
| | 2.3 | | ty population | |
| 2 | Dline | | | |
| 3 | Biind | iea re | eview of the data | 12 |
| 4 | Stati | stical | and analytical methods | 13 |
| | 4.1 | Gen | eral statistical considerations | 13 |
| | 4.2 | Miss | sing data handling | 13 |
| | 4.3 | Base | eline definition | 14 |
| | 4.4 | Defi | nition of study visit and visit window | 15 |
| | 4.4. | .1 | Study visit | |
| | 4.4. | .2 | Visit window | 15 |
| | 4.5 | Pati | ent disposition | 15 |
| | 4.6 | Den | nographics and baseline characteristics | 15 |
| | 4.7 | Med | dical history | 15 |
| | 4.8 | Ben | efit analyses | 16 |
| | 4.8. | | Primary analyses | |
| | 4.8. | .2 | Secondary analyses | 17 |
| | 4.9 | Safe | ty analyses | 17 |
| | 4.9. | .1 | Primary analyses | 17 |
| | 4.10 | Mod | deling and estimating | 18 |
| | 4.10 | 0.1 | Model and statistical test for the effect of treatment on DAS28 (Hypotheses 1) | 18 |

| | 4.10 | 0.2 | Model and statistical test for the effect of treatment on damage score (hypothesis | 2) |
|---|---|---|---|---|
| | | | | 21 |
| | 4.10 | 0.3 | Model and statistical test for the effect of treatment on harm: SAEs or other AESIs (Hypotheses 3) | . 22 |
| | 4.11 | Eval | uation of possible confounded results due to differential co-intervention | 22 |
| | 4.13 | 1.1 | Testing and correcting for differential treatment changes | 23 |
| | 4.12 | Inte | rpretation rules | 25 |
| | 4.13 | Anal | ysis of secondary outcome variables | 26 |
| 5 | Inter | im ar | nalyses | 27 |
| 6 | Samı | ole siz | ze and power calculations | 27 |
| 7 | Table | es, lis | tings and figures | 29 |
| 8 | Stati | stical | software | 76 |
| 9 | Refe | rence | S | 76 |
| 10 | Арре | endix | A: secondary outcome measures that need further specification | 78 |
| 11 | Арре | endix | B – Modifications from the protocol | 80 |
| 12 | Арре | endix | C. Report of blinded data review meetings | 82 |
| | Appe | | D. Gloria final PP population, also excluding initial changes in antirheumatic | 85 |

## List of abbreviations and definitions

| aCCP | Anti-CCP |
|---|---|
| ACR | American College of Rheumatology |
| AE | Adverse event |
| AESI | Adverse event of special interest |
| CI | Confidence Interval |
| CRP | C-reactive protein |
| DAS | Disease activity score |
| DEXA | Dual-energy X-ray absorptiometry |
| DMARD | Disease-modifying antirheumatic drugs |
| ESR | Erythrocyte sedimentation rate |
| EULAR | European League Against Rheumatism |
| EQ-5D | Euro-QoL in 5 dimensions |
| GC | Glucocorticoid |
| GCP | Good Clinical Practice |
| GLORIA | The Glucocorticoid Low-dose Outcome in Rheumatold Arthritis Study |
| GRADE | Grades of Recommendations, Assessment, Development, and Evaluation |
| GTI | Glucocorticoid Toxicity Index |
| HAQ | Health Assessment Questionnaire |
| ITT | Intent-to-treat |
| LRT | Log-likelihood-ratio test |
| MAR | Missing at random |
| MCAR | Missing completely at random |
| MDA | Minimal disease activity |
| MICE | Multiple imputation by chained equations |
| NMAR | Not missing at random |
| NSAID | Non-steroidal anti-inflammatory drug |
| PP | Per protocol |
| QALY | Quality-adjusted life years |
| QoL | Quality of life |
| RA | Rheumatoid arthritis |
| RAID | RA Impact of Disease |
| RF | Rheumatoid factor |
| SAE | Serious adverse event |
| SAF | Safety |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SDAI | Simple Disease Activity Index |
| SF-36 | Short Form 36-item Health Survey |
| WHO-ILAR | World Health Organisation/International League of Associations for |
| | Rheumatology |

#### 1 Introduction

We present the analysis plan executed on the data collected according to the GLORIA protocol. The analysis plan summarizes the study protocol, describes the statistical methods, data listings and summary tables for the analysis of the data from the GLORIA trial. Any differences with the original protocol will be documented.

The details of the economic evaluation and analysis of the adherence substudy will be described in a separate analysis plan.

#### 1.1 Study population

The study population consists of patients of 65 years or older with rheumatoid arthritis (RA) according to the 1987 or 2010 classification criteria of the American College of Rheumatology (ACR) and the European League Against Rheumatism (EULAR) (Aletaha, 2010), requiring antirheumatic therapy because of inadequate disease control, as evidenced by a 28-joint disease activity score (DAS28) of ≥2.60. Patients were selected from 28 hospitals in Germany, Hungary, Italy, The Netherlands, Portugal, Romania and Slovakia.

#### 1.2 Study design

The GLORIA study is a randomized, double-blind, placebo-controlled pragmatic multicenter clinical trial to assess the effectiveness and safety of a daily dose of 5 mg prednisolone or matching placebo in elderly RA patients. Patients will be randomized into two arms: the experimental arm (receiving prednisolone 5 mg/day) or the control arm (receiving placebo). The trial period is 24 months with 3 additional months during which study medication treatment is tapered. In the first 3 months, comedication is limited: co-medication can be changed only at baseline or after 3 months, creating a brief period in which the effects of prednisolone can be studied with minimum interference.

Our design emulates the routine care setting: eligibility criteria are minimal, assessments and procedures are tailored to represent standard of care, and concurrent antirheumatic treatment is allowed next to the trial medication with minimal limitations. Thus we expect that almost all elderly RA patients (specifically those with comorbidities) are eligible.

The adherence of all patients in the main GLORIA trial is monitored throughout the study period by an adherence monitoring device loaded into the cap of the drug bottle, and by a count of returned capsules at every clinic visit.

Assessment takes place at varying intervals and includes 7 clinic visits and 3 assessments by telephone. The sequence and duration of all study periods is represented in Figure 1.

Figure 1: Schedule of assessments

| | Base<br>-line | | | 2 | year trea | itment pe | riod | | | Follow-<br>up /<br>taper |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit No | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| Month (visit window +/- 2 months) | 0 | 3 | 6 | 9 | 12 | 15 | 18 | 21 | 24 <sup>LV</sup> | 27 |
| Location | clinic | clinic | clinic | remot<br>e | clinic | remot<br>e | clinic | remot<br>e | clinic | clinic |
| Written informed consent | Х | | | | | | | | | |
| In- / exclusion criteria | Х | | | | | | | | | |
| Demographics, education & medical history | Х | | | | | | | | | |
| Baseline prognostic factors:<br>adherence, health literacy, arthritis<br>helplessness index | X* | | | | | | | | | |
| Randomization | X* | | | | | | | | | |
| Physical examination | Х | | | | | | | | | |
| Height | Х | | | | | | | | Х | |
| Vital signs / weight | Х | Х | Х | | Х | | Х | | Х | Х |
| AE evaluation (inc. surgery, comorbidity) (safety) | | X* | X* | X* | X* | X* | X* | X* | X* | X* |
| Concomitant medication | X | X | Х | Х | Х | Х | Х | X | Х | Х |
| Lab (hematology <sup>1</sup> , chemistry <sup>2</sup> ) | Х | Х | Х | | Х | | Х | | Х | |
| Lab lipids <sup>3</sup> | X | X | | | X <sup>3</sup> | | | | Х | |
| Lab CRP, ESR | X | X | Х | | Х | | Х | | Х | Х |
| Joint counts (44) (effectiveness) | X | | | | | | | | Х | |
| Joint counts (28) (effectiveness) | | X | Х | | Х | | Х | | | Х |
| DEXA either with VFA,<br>or without VFA plus<br>X-lat spine (thor, lumb) <sup>4,5</sup> | Х | | | | | | | | Х | |
| X-rays hand and forefeet <sup>4</sup> (safety) | X | | | | | | | | Х | |
| Patient global assessment, stiffness duration, stiffness severity | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Physician global assessment | X | X | Х | | Х | | Х | | Х | Х |
| Questionnaires: | | | | | | | | | | |
| - RAID | X* | X* | X* | X* | X* | X* | X* | X* | X* | X* |
| - full HAQ-DI (24 items) | X* | X* | X* | | X* | | X* | | X* | X* |
| - MHAQ-DI (10 items) | | | | X | | X | | X | | |
| - Cost questionnaire | X* | X* | X* | | X* | | X* | | X* | X* |
| - EQ-5D | X* | X* | X* | X* | X* | X* | X* | X* | X* | X* |
| - SF36 | X* | | | | | | | | X* | |
| - Patient symptom list | X* | | | | | | | | X* | X* |
| GC or placebo, dispense adherence | X* | X* | X* | X* | X* | X* | X* | X* | X* | |

<sup>\*</sup> procedures not belonging to standard of care

Iv End of study visit. This visit also needs to be completed by subjects who early terminated the trial.

Apart from CRP and ESR, the following standard of care lab tests will be done on peripheral blood samples.

Lab results of CRP and ESR no more than 4 weeks old may be used for the baseline visit.

Results of the below tests 1,2,3 no more than 2 months old may be used for the baseline visit:

- 1) Hemoglobin, Mean Cell Volume, White blood cell count, White blood cell differential count, Platelet count.
- 2) Glucose (non-fasting), Creatinine, Alanine Aminotransferase;
- 3) Total cholesterol, HDL cholesterol. Optional for month 12.
- 4) For the baseline visit: DEXA, DEXA VFA and X-ray images with a maximum of 6 months before or until 3 months after the baseline visit may be used.
- 5) If possible a whole body DEXA may be performed.

#### 1.3 Primary and secondary study objectives

#### 1.3.1 Primary objectives

The primary objectives of the GLORIA project are to compare the effect of low-dose GC therapy (5 mg/day), relative to placebo, on time-averaged mean value of the disease activity *AND* the number of patients experiencing at least one AE of Special Interest for two years as co-treatment in elderly RA patients ( $\geq$ 65 years).

#### 1.3.2 Secondary objectives

- To assess study medication adherence through a medication packaging solution; and, in a substudy, test the effectiveness of smart device technology to improve adherence (separate statistical analysis plan, not described here).
- To assess the secondary outcome measures which are described in section 1.4.2.
- Deliver an outcome prediction model for individual patient outcome, to tailor treatment strategies for elderly RA patients with comorbidities
- Deliver data to support:
  - Better guidelines on RA treatment in elderly
  - More accurate information for elderly RA patients, their physicians and researchers
  - Improved strategies for trial design and conduct in the elderly

#### 1.4 Primary and secondary endpoints

#### 1.4.1 Primary endpoints

- To measure benefit, the primary endpoints are:
- a) signs and symptoms: the time-averaged mean value (estimated from linear mixed models) of the DAS28;
- b) damage score: change from baseline after 2-years in total Sharp/van der Heijde damage score of hands and forefeet radiographs.
- To measure safety, the primary endpoint is the total number of patients experiencing at least one adverse event of Special Interest (AESI). An AESI is defined as either a serious adverse event (SAE) according to the GCP definition, or the occurrence of one of the following AEs ('other AESI'):
  - Any AE (except loss of efficacy, worsening of disease) that leads to the definite cessation of the trial medication;
  - A cardiovascular event (myocardial infarction, cerebrovascular event, peripheral arterial vascular event);
    - Anything falling outside this definition is not an AESI.

      So venous hemorrhoids, venous ulcus cruris, thrombosis, pulmonary embolism, subdural hematoma, and traumatic hemorrhagic brain lesions are not coded as AESI. Also cardiac rhythm disturbances, valve lesions, cardiac insufficiency, cardiomyopathy, and encephalopathy, are not coded as AESI unless part of an acute ischemic episode.
  - Newly occurring hypertension requiring drug treatment;

- Newly occurring diabetes mellitus requiring drug treatment;
- Symptomatic bone fracture requiring treatment;
  - AESI is coded as 'no' if the vertebral fracture was asymptomatic, and 'yes' for all nonvertebral fractures, unless expressly indicated that the fracture was asymptomatic.
    - Note that vertebral fracture is also captured as secondary outcome through DEXA or spine radiographs.
- o Infection requiring antibiotic treatment;
  - Any specific treatment aimed at microorganisms to treat an infection is included: includes topical, antiviral, antifungal, antiparasitic treatment.
  - (Surgical) procedures with concomitant antibiotics: not (initially) an infection, so not AESI; AESI only when the procedure was done for a primary infection (e.g. abscess). Surgical complications treated with antibiotics are also not coded as AESI, because it is usually impossible to determine whether the antibiotic was given as prophylaxis or as treatment.
    - Note: almost any surgery is of necessity (hospital admission) already an SAE.
- Newly occurring cataract or glaucoma.
  - Cataract and glaucoma are assumed to be bilateral. A medical history of the disease in one eye counts for both, so no AESI during the trial for procedures on the contralateral eye. We count bilateral procedures for new disease as one (not two) AESI.

AEs can be reported spontaneously by patients, on prompting at clinic visits or by telephone interviews, and by the treating physician. The AEs specified above will be recorded with special care in a separate procedure. This procedure includes adjudication through the collection of evidence. This can be a declaration of the treating physician (in case of start of treatment, or a copy of a letter confirming the event, kept on file in the center.

The safety database uses the regular term and definition to describe SAE. The electronic Case Record Form and study database uses AESI to describe events that match one of the other bullets, regardless of whether the event is an SAE. So there an event can be labeled SAE (y/n) and separately AESI (y/n). In the primary analysis patients will be counted who have at least one SAE or AESI as scored in the safety database ('other AESI'), to match with the definition of primary endpoint specified above.

From here, the primary endpoint for safety is defined as 'SAE or other AESI' because one AE can be labeled as a SAE as well as an AESI.

- Cost-effectiveness and cost-utility: more details are described in the separate analysis plan for the cost analyses
- Medication adherence: adherence to trial drug is measured through the e-communicative packaging solution as the count of days in which the bottle is opened on the appropriate days, as measured by the adherence tool. The tool (cap) is collected during the study visits at 3, 6, 12, 18, 24 and 27 months. Each cap is sent back to the provider and the data are read out centrally.

#### 1.4.2 Secondary endpoints

#### Benefit

- WHO-ILAR core set of RA outcome measures, including patient and physician global assessment of disease activity, joint counts (swollen joints and tender joints), acute phase reactants (C-reactive protein (CRP) and erythrocyte sedimentation rate (ESR)) at 0, 3, 6, 12, 18, 24 and 27 months, and radiographs of hands and forefeet at 0 and 2 years.
   Remaining core set measures: pain and fatigue are part of the RAID questionnaire (see below), and physical function is assessed by the (m)HAQ.
- DAS44 at 0 and 24 months
- DAS28 at 3, 6, 12, 18, and 27 months
- Severity and duration of morning stiffness at every study visit
- SF36 The Short Form 36-item Health Survey, a questionnaire about quality of life (QoL) at 0 and 24 months
- 57-symptom list at 0 and 24 months
- RA Impact of Disease (RAID) tool The RAID is a validated questionnaire assessing the seven
  most important domains of impact of RA on the patients: pain, functional disability
  assessment, fatigue, sleep, physical well-being, emotional well-being, coping. at every
  study visit
- (Modified) Health Assessment Questionnaire ((m)HAQ) at every study visit
- RAPID3, calculated with the patient global assessment of disease activity, (m)HAQ and the question about pain from the RAID questionnaire, at every study visit
- Cost questionnaire at 0, 3, 6, 12, 18, 24, 27 months, including
  - Activity limitation
  - Work disability (for those holding a paid job)
- Utility/Quality-adjusted life years (QALY): Euro-QoL in 5 dimensions (EQ-5D) at every study visit

#### Harm

- Vital signs (heart rate and blood pressure), height, weight at 0, 3, 6, 12, 18, 24, 27 months
- Bone mass assessed by Dual-energy X-ray Absorptiometry (DEXA) at 0 and 24 months
- Vertebral Fracture Analysis (by DEXA OR lateral radiograph of thoracic and lumbar spine) at 0 and 24 months
- Discontinuation of study drug with reason: this includes patients in whom treatment with prednisolone becomes clinically indicated or those with unacceptable side effects attributable to study medication
- Change of antirheumatic treatment, with reason
- Intensification of treatment for existing comorbidity, e.g. hypertension or diabetes
- Joint replacement surgery
- AEs, SAEs, other AESI at every study visit
- Concomitant medication at every study visit

Data collection is in agreement with industry standard (i.e. Meddra terminology etc.).

#### GC harm/benefit balance

Blood samples will be collected during the study as part of the standard of care of RA patients, of which non fasting blood samples at 0, 3, 6, 12, 18, 24 and 27 months. No additional blood samples will be taken for this study. In specific cases, extra lipid analysis will be performed on the blood samples collected as part of the standard of care.

#### Medication adherence

• Adherence to the trial drug is measured through the e-communicative packaging solution as the count of days in which the bottle is opened on the appropriate days (pill count), as measured by the adherence tool at 3, 6, 12, 18, 24 and 27 months

#### Other

- Demographics, education and medical history at baseline
- Baseline prognostic factors: Morisky medication adherence scale (MMAS-8), health literacy, arthritis helplessness index questionnaires at baseline
- Cost-effectiveness and cost-utility: estimate of costs of treatment and monitoring
- Patients retained on study drug over time: survival analysis

#### 2 Analysis populations

For the full trial period, we will perform analyses of the primary and secondary outcome variables on the intent-to-treat (ITT) population, with ad-hoc sensitivity analyses excluding selected patients based on blinded data review. The ITT principle asserts the effect of a treatment policy (that is, the planned treatment regimen), rather than the actual treatment given (i.e., it is independent of treatment adherence etc.). Accordingly, participants allocated to a treatment group (GC and placebo, respectively) should be followed up, assessed and analysed as members of that group, irrespective of their adherence to the planned course of treatment (i.e., independent of withdrawals and cross-over phenomena). Primary safety analyses will be repeated in the safety (SAF) population.

#### 2.1 Intent-to-treat population

The intent-to-treat population is defined for efficacy as all patients randomized into the study who took the study medication (prednisolone or placebo) for at least one day and who have at least one baseline and one follow-up assessment. Patients will be analyzed in the group they were randomized to.

# 2.2 Per-protocol population, also excluding initial changes in antirheumatic medication

For the 3-month efficacy assessment: this population consists of all patients who during the first 3 months:

- received the study drug;
- had at least 80% adherence to treatment as determined by tablet count;
- completed the baseline and 3-month visit;
- have a DAS28ESR value available on both visits; or a DAS28CRP value on both visits;
- did not start, stop or change the dose of concurrent antirheumatic drugs, or receive glucocorticoid (oral or injection) at baseline or in the period up to the 3-month visit:
- did not have any serious protocol violations as determined in section 3.

The report from the blinded data review and the list of patients excluded from this population have finalized before the database is locked and are attached to this plan (appendix C).

#### 2.3 Safety population

All patients who took at least one capsule of study medication belong to the safety population.

#### 3 Blinded review of the data

Multiple blinded data review meetings with the principal investigator, medical monitor, study lead, trial statistician, a representative of data management and a member of the scientific advisory committee will be held before breaking the blind. During the blinded data review the protocol violations and their impact on the study outcomes will be discussed. The decisions taken during the blinded data review will be finalized and signed by the participants of this meeting before breaking the blind. The final report of these meetings are attached as appendix C.

### 4 Statistical and analytical methods

#### 4.1 General statistical considerations

All continuous variables will be summarized with the following descriptive statistics: number of patients (n), mean, standard deviation (SD). If the data are non-normally distributed, median, minimum (min.) and maximum (max.) will be reported. For categorical variables, the absolute (N) and relative frequency (%) will be reported.

#### 4.2 Missing data handling

Handling of missing DAS28 (disease activity) outcomes (applies to DAS28-ESR and DAS28-CRP)
Step 1. Imputation of missing DAS28 if only the component 'patient global assessment of disease activity' is missing

If the missing DAS28 score is from an intermediate (i.e. not baseline or end) visit and only the patient global assessment of disease activity is missing, it will be replaced by the mean of the patient global score immediately before and after this visit, and the DAS28 score will be calculated with this result. If one or both of these are also missing the value will remain missing because we have no information to impute a value.

Step 2. All remaining missing DAS28

In principle, DAS28 outcomes may be incomplete for two reasons:

- 1. Non-monotone missingness, for example because a patient skips a clinic visit/measurement occasion but is observed again at later points in time
- 2. Monotone missingness in case of premature discontinuation of study medication

For the primary analysis, we use single imputation by chained equations using the MICE package (van Buuren 2012) to impute missing values according to the following rules. At each study time point we observe or do not observe patient's DAS28, DAS28-CRP, and RAPID-3 score. We impute missing values on these variables per measurement occasion, if at least one measurement is present. If all three measurements are missing, we do not impute any value. These cases usually occur due to discontinuation of the study. The main analysis model (section 4.10) is a mixed effects longitudinal model which gives consistent estimates under the assumption that the remaining missing DAS28 outcomes are missing at random (Little and Rubin 2002).

Sensitivity analysis: Nonresponder imputation

Finally, in case of monotone missingness we investigate the possibility that the missingness occurs not at random (NMAR) with robustness analyses (nonresponder imputation). This imputation method recodes the outcomes of all complete units observed at the end of the study period (j=m),  $Y_m$ , as follows:

$$\tilde{Y}_m = \begin{cases} 1 & iff \ Y_m - Y_1 < 0.6 \\ 0 & iff \ Y_m - Y_1 \ge 0.6 \end{cases}$$

where 0.6 denotes a minimum effect. Incomplete units receive  $\tilde{Y}_m = 0$  representing the conservative hypothesis that all incomplete cases would not have achieved a minimum treatment effect.

Subsequently, we test whether the proportions of responders ( $\tilde{Y}_m = 1$ ) differs significantly between treatment and placebo with a model for difference in proportions akin to model 3 in section 3.3.

#### Handling of missing damage scores

Step 1. Handling of assessments with partially missing data

Joints with signs of surgery (e.g. prosthesis, arthrodesis) are not scored. Also, when assessments at both time points have been done, but groups of joints are missing from one time point, the scores from that group are also set to missing at the other time point. For example if the end assessment includes only hand films (feet films missing), the initial assessment of the feet will be set to missing. Likewise, if surgery is done on a joint during the trial, the initial assessment of that joint will also be set to missing.

#### Step 2. All remaining missing damage assessments

We may distinguish three missing data patterns in the damage scores at study onset and study endpoint:

- 1. Damage score is not observed at study onset but the endpoint is observed,
- 2. Damage score is observed at study onset but the endpoint is unobserved,
- 3. Damage score is neither observed at study onset nor endpoint.

The three missing data patterns are addressed as follows.

For the primary analysis, we use the algorithm 'MICE' (multiple imputation by chained equations) to impute missing measurements (van Buuren, 2012). This procedure assumes missing at random (MAR) data. The imputation models use data available at baseline (damage score at baseline, disease duration, rheumatoid factor positivity, ACPA positivity, DAS28-ESR) and the endpoint measurement of damage. Study center is not taken into account in this imputation model in view of the large number of cases with missing endpoints.

As a sensitivity analysis, we conduct a complete case analysis deleting all cases with (remaining) missing onset outcomes or missing endpoint outcomes list-wise. This analysis thus excludes cases with patterns 1, 2 and 3. This analysis assumes these outcomes are missing completely at random, MCAR (Little & Rubin, 2002).

#### Handling of missing harm outcomes

Harm is verified throughout the trial via remote and onsite checks against the source data. So harm assessment is assumed to be complete.

#### 4.3 Baseline definition

Baseline is defined as the last value immediately before the start of the treatment.

#### 4.4 Definition of study visit and visit window

#### 4.4.1 Study visit

The baseline visit (visit 1, in the clinic) is defined as study month 0. The next visits are at 3 months (visit 2, in clinic), 6 months (visit 3, in clinic), 9 months (visit 4, remote), 12 months (visit 5, in clinic), 15 months (visit 6, remote), 18 months (visit 7, in clinic), 21 months (visit 8, remote), 24 months (visit 9, in clinic), 27 months (10, in clinic). The end of the study is defined as the date of the last study visit.

#### 4.4.2 Visit window

The protocol allowed to minimize or maximize the visit window with two months. For the radiology data (x-rays hand and forefeet and DEXA), the time window for the baseline measurement was 6 months before or 3 months after the baseline visit, and for the 24-months measurement 3 months before or after visit 9. If these are exceeded we will accept images up to 1 year before and 6 months after baseline, and up to 1 years after year 2. Data will be analyzed based on the visit number/month that is reported in the database. The calendar visit dates will not be used.

#### 4.5 Patient disposition

The number and percentages of patients allocated to the prednisolone and placebo group will be summarized for all enrolled patients. The number and percentage of patients completing and withdrawing the study, the reasons of withdrawal, and study duration will be reported in a table overall and by treatment.

#### 4.6 Demographics and baseline characteristics

Demographics and baseline characteristics, including birth month and year, sex, smoking, alcohol use, the possession of a smartphone, education level, rheumatoid factor (RF) status, anti-CCP (aCCP) status, duration of RA, evidence of structural joint damage, previous related surgical procedures, previous glucocorticoid use, previous NSAID use, previous DMARD use, previous biological use, number of comorbidities will be reported in a table by treatment group and overall.

#### 4.7 Medical history

Number and percentages of patients with a history of diseases, abnormalities or surgery will be summarized by treatment group and overall. The reported term, preferred term, system organ class, and year of resolution or ongoing will be listed. The MedDRA coding dictionary, version 21.0, will be used to code the medical history.

#### 4.8 Benefit analyses

#### 4.8.1 Primary analyses

#### 4.8.1.1 DAS28

The following primary benefit hypotheses will be tested for the DAS28 score:

1a. Primary benefit hypotheses:

 $H_{0,1a}$ : (Null) Prednisolone intake over a period of 24 months leads on average to no difference or a higher score in DAS28 than placebo intake.

 $H_{1,1a}$ : (Alternate) Prednisolone intake over a period of 24 months leads on average to a lower score in DAS28 than placebo intake.

$$H_{0.1a}$$
:  $\mu_{\rm T}(t=24) - \mu_{\rm C}(t=24) \ge 0$ 

$$H_{1.1a}$$
:  $\mu_{\rm T}(t=24) - \mu_{\rm C}(t=24) < 0$ 

 $\mu_T(t=24)$  is the mean of DAS28 over 24 months in the treatment group.  $\mu_C(t=24)$  is the mean of DAS28 over 24 months in the control group.

#### 4.8.1.2 Damage score/progression

Damage progression is analyzed as damage at end, with baseline damage as covariate (see model, section 4.10).

The following primary benefit hypothesis will be tested for damage:

2a. Primary benefit hypothesis:

H<sub>0,2a</sub>: (Null) Prednisolone intake over a period of 24 months leads on average to no difference or a higher damage progression compared to placebo intake.

H<sub>1,2a</sub>: (Alternate) Prednisolone intake over a period of 24 months leads on average to a lower damage progression compared to placebo intake.

$$H_{0.2}$$
:  $\delta_{\rm T}(t=24) - \delta_{\rm C}(t=24) \ge 0$ 

$$H_{1,2}$$
:  $\delta_{\rm T}(t=24) - \delta_{\rm C}(t=24) < 0$ 

 $\delta_T(t=24)$  is the mean damage score at 24 months in the treatment group.  $\delta_C(t=24)$  is the mean damage score at 24 months in the control group.

#### 4.8.2 Secondary analyses

The following secondary benefit hypothesis will be tested for the DAS28 in the per-protocol population (see 2.2):

1b. Secondary benefit hypotheses:

 $H_{0,1b}$ : (Null) Prednisolone intake over a period of 3 months leads on average to no difference or a larger score in DAS28 than placebo intake.

 $H_{1,1b}$ : (Alternate) Prednisolone intake over a period of 3 months leads on average to a smaller score in DAS28 than placebo intake.

$$H_{0.1b}$$
:  $\mu_{\rm T}(t=3) - \mu_{\rm C}(t=3) \ge 0$ 

$$H_{1,1b}$$
:  $\mu_{\rm T}(t=3) - \mu_{\rm C}(t=3) < 0$ 

#### 4.9 Safety analyses

#### 4.9.1 Primary analyses

The following primary harm hypothesis will be tested:

*3a. Primary harm null hypothesis:* 

 $H_{0,3a}$ : (Null) The probability of patients receiving prednisolone to encounter at least one SAE or other AESI (as defined in the protocol) in a period of 24 months is equal to or less than the probability of patients receiving placebo.

 $H_{1,3a}$ : (Alternate) The probability of patients receiving prednisolone to encounter at least one SAE or other AESI in a period of 24 months is greater than the probability of patients receiving placebo.

$$H_{0.3a}$$
:  $\pi_{\rm T}(t=24)/\pi_{\rm C}(t=24) \le 1$ 

$$H_{1,3a}$$
:  $\pi_{\rm T}(t=24)/\pi_{\rm C}(t=24) > 1$ 

 $\pi_T(t=24)$  is the probability to encounter an SAE or other AESI over a 24 months period in the treatment group.  $\pi_C(t=24)$  is the probability to encounter an SAE or other AESI over a 24 months period in the control group.

#### 4.10 Modeling and estimating

The testing of the hypothesis sets requires estimating the average effect of treatment on benefit (operationalized as DAS28 and progression of joint damage) and harm (operationalized as encountering at least one SAE or other AESI). An observed effect with a probability of occurrence under the (one-sided) null hypothesis (p-value) of 5% or less will be considered significant causing us to reject the null and to accept the alternative hypothesis. The hypotheses and their tests are one-sided in view of pre-existing knowledge for benefit and the likelihood that true benefit will be underestimated in the context of the pragmatic design and potential differential co-intervention (see section 4.11); and for harm because of limited power. This results in a higher chance of declaring benefit, but also a higher chance of declaring harm.

The average effect of treatment on DAS28 (hypotheses 1) and damage progression (hypothesis 2) will be estimated in a mixed effects regression model. The exact form and empirical fit of the model are important determinants of the power of the statistical test of the treatment effect parameter, as described below. Hypotheses 3 require estimation of the difference in probability to encounter a SAE or other AESI between treatment and placebo over 24 months, which will be implemented by estimating the odds ratio of a SAE or other AESI in treatment versus placebo. All analyses will also take into account that the GLORIA study uses a stratified sampling design, where within each of 28 participating centers randomization is executed stratified by earlier exposure to glucocorticoids (yes/no) and start or switch of other anti-rheumatic drugs at the beginning of the trial.

We first describe how hypothesis testing for the GLORIA study will be executed. In this exposition, we assume that the observed data matrix is complete and that the estimated effects are not confounded with treatment changes. We describe methods to address incomplete data (section 4.2) and to assess confounding with treatment changes (section 4.11).

Our general analysis strategy can be summarized as follows:

- 1. Test hypotheses 1 to 3 with models described in this section and missing-at-random data correction (section 4.2).
- 2. Execute robustness checks for monotonous not-missing-at-random data pattern with non-responder imputation (NRI; section 4.2).
- 3. Assess confounding with treatment changes (section 4.11)
- 4. Formulate rules to interpret the overall trial results (section 4.12)

#### 4.10.1 Model and statistical test for the effect of treatment on DAS28 (Hypotheses 1)

We first consider the analysis of the DAS28 outcome (benefit). The measurement level of DAS28 may be considered continuous so that we can model outcomes by continuous variable models. In the analysis, we need to solve two problems: first, how to estimate an average effect across the study period of two years, and second, how to take the longitudinal data structure into account. The second aspect poses two sub-problems; first, whether to treat time as continuous or discrete and, second, how to take into account that repeated measurements on the same individual are correlated (standard regression techniques assume uncorrelated observations).

The problem of intra-individual correlated observations will be addressed by mixed-effect regression models. The primary distinction in mixed-effect models for longitudinal data is the treatment of time in the model. In so-called fixed-occasion designs, time takes on a discrete form, whereas in so-called variable-occasion designs time takes on a continuous form (Hox, 2010; Snijders & Bosker, 2011). Fixed occasion designs are characterized by the fact that at given occasions outcomes of all (or most) of subjects are observed. Variable occasion designs are not limited by this restriction and there may be a large number of occasions at which only few subjects need to be observed.

Although the design of the GLORIA study in principle lends itself to both types of model classes we will test hypotheses 1 with a fixed occasion model, because the number of time points at which individuals are observed is limited (up to six) and the model can accommodate non-linear trends in the data well by including occasion specific effects and occasion-treatment interactions (see expectations in figure 2). Continuous time models may also accommodate non-linear trends, but then the specification of the functional form becomes crucial and we do not have strong prior expectations of any particular functional model. We note continuous time models may be considered for secondary analyses.

#### 4.10.1.1 Full model

We model the treatment outcome by a mixed effect model with fixed effects measurement occasion after baseline (d), baseline measurement (Z), treatment condition (T), and random effects across individuals (level 2; random intercept U) and study centers (level 3; random intercept V). Furthermore, we include the strata of the GLORIA trial (S) as fixed effects. Centers could also be modeled as fixed effects, but we have chosen random effects because several centers have included only a very low number of patients. A compound symmetry correlation structure is assumed.

We write down mixed effect model 1 as:

```
Y_{ijk} = \beta_{0jk} + \sum_{s=1}^{4} \beta_{1jks} d_{ijks} + \epsilon_{ijk}
                                                                                                            (level-1 model)
\beta_{0ik} = \delta_{00k} + \delta_{01k}S_{ik1} + \delta_{02k}S_{ik2} + \delta_{03k}T_{ik} + \delta_{04k}Z_{ik} + U_{0ik}
                                                                                                            (level-2 model for intercept)
\beta_{1iks} = \delta_{10ks}
                                                                                                            (level-2 model for slope)
\delta_{00k} = \gamma_{000} + V_{00k}
                                                                                                            (level-3 model for intercept)
\delta_{01k} = \gamma_{010}
                                                                                                            (level-3 model for slope)
                                                                                                            (level-3 model for slope)
\delta_{02k} = \gamma_{020}
                                                                                                            (level-3 model for slope)
\delta_{03k} = \gamma_{030}
                                                                                                            (level-3 model for slope)
\delta_{04k} = \gamma_{040}
                                                                                                            (level-3 model for slope)
\delta_{10ks} = \gamma_{100s}
```

with  $U_{0jk}$  the individual-level random effect,  $V_{00k}$  the center-level random effect, and  $\epsilon_{ijk}$  the residual.

#### The indices:

i= 1,..., m: fixed measurement occasion after baseline (in GLORIA, m=5)

j= 1,...,n: individuals

k=1,...,K: study centers (currently, K=28 in GLORIA)

#### The variables:

 $Y_{ijk}$ : DAS28 outcome

 $d_{ijks}$ : dummy variables encoding the five measurement occasions after baseline, s=1,..., 4

 $T_{jk}$ : treatment indicator, 0 if placebo, 1 if active (prednisolone) treatment

 $Z_{ik}$ : Baseline measurement of DAS28

 $S_{ik1}$ ,  $S_{ik2}$ : Stratification factors

#### The parameters:

 $\gamma_{000}$ : the model intercept

 $\gamma_{010}$ : fixed effect of stratification factor 1  $\gamma_{020}$ : fixed effect of stratification factor 2

 $\gamma_{030}$ : fixed effect of treatment

 $\gamma_{040}$ : fixed effect of baseline measurement of DAS28

 $\gamma_{100s}$ : effect of time dummy s

#### And the random effects:

 $U_{0jk}$ : random intercept of individual i  $V_{00k}$ : random intercept of study center

 $\epsilon_{iik}$ : residual

In hypotheses 1, we test for a difference in mean DAS score across a time of 24 months between treatment and placebo. In model (1), this difference in means is estimated by parameter  $\gamma_{030}$ . For the PP analysis at 3 months, the model becomes two-level (no time) as there is only one assessment post baseline.

#### 4.10.1.2 Testing and exploration of treatment-time interactions

The significance of all parameters in model 1 is evaluated using t-tests with Satterthwaite's method for approximating degrees of freedom (Kuznetsova, Brockhoff, and Christensen, 2017). In particular, hypothesis H1a is tested by evaluating the one-sided p-value of  $\gamma_{030}$  rejecting the one-sided null hypotheses if  $\gamma_{030} < 0$  significantly and not rejecting else. The main effect of measurement occasions across all dummy variable d is evaluated jointly by a likelihood ratio test (LRT).

After this assessment, we will explore in a secondary analysis if the interaction between treatment and measurement occasions (time) interaction is significant using a LRT. If this test is significant we will test at which measurement occasions there is a significant difference using t-tests with Bonferroni correction of the p-values.

#### 4.10.2 Model and statistical test for the effect of treatment on damage score (hypothesis 2)

The treatment effect on the damage score at 24 months (hypothesis 2) will be evaluated by the total Sharp/van der Heijde damage score of hands and forefeet. We will use a linear mixed-effects regression model defined similarly to model 1. Contrary to model 1 there are no repeated measurements. Therefore, we model outcomes of individuals nested in centers and include as main effects treatment, design strata, and the baseline measurement of the damage score. A random effect for study center is included. Model 2 is formalized as follows:

| $Y_{jk} = \delta_{0k} + \delta_{1k} S_{jk1} + \delta_{2k} S_{jk2} + \delta_{3k} T_{jk} + \delta_{4k} Z_{jk} + U_{jk}$ | (level-1 model) |
|---|---|
| $\delta_{0k} = \gamma_{00} + V_{0k}$ | (level-2 model for intercept) |
| $\delta_{1k} = \gamma_{10}$ | (level-2 model for slope) |
| $\delta_{2k} = \gamma_{20}$ | (level-2 model for slope) |
| $\delta_{3k} = \gamma_{30}$ | (level-2 model for slope) |
| $\delta_{4k} = \gamma_{40}$ | (level-2 model for slope) |

where now  $Y_{jk}$  is the damage score at 24 months and  $Z_{jk}$  is the damage score at baseline. Equivalent to section 3.1.1, it can be see that if a one-sided t-test of  $\gamma_{30} < 0$  is significant,  $H_{0.2}$  is rejected.

We note that the damage progression measurement can be positively skewed, threatening the accuracy (type 1 error rate) of the statistical tests in small samples (and other tests of regression coefficients including t- and F-tests). If we observe a strongly skewed distribution we will apply a bootstrapped test procedure instead of the t-test.

# 4.10.3 Model and statistical test for the effect of treatment on harm: SAEs or other AESIs (Hypotheses 3)

Contrary to the hypothesis set 1 on the benefit of prednisolone treatment, hypotheses 3 require testing the difference in probabilities of encountering at least one SAE or other AESI over 24 months. On marginal level it would be sufficient to estimate these probabilities after t=24 months and evaluate the significance of their difference. However, to additionally account for the stratification of the GLORIA design, we apply a logistic mixed-effects regression (model 3):

$$P_{jk} = g^{-1}(\delta_{0k} + \delta_{1k}S_{jk1} + \delta_{2k}S_{jk2} + \delta_{3k}T_{jk} + U_{jk})$$

| $\delta_{0k} = \gamma_{00} + V_{0k}$ | (level-2 model for intercept) |
|--------------------------------------|-------------------------------|
| $\delta_{1k} = \gamma_{10}$ | (level-2 model for slope) |
| $\delta_{2k} = \gamma_{20}$ | (level-2 model for slope) |
| $\delta_{3k} = \gamma_{30}$ | (level-2 model for slope) |
| $\delta_{4k} = \gamma_{40}$ | (level-2 model for slope) |

where now  $P_{jk}$  the probability of patient j in center k to encounter at least one SAE or other AESI over 24 months. The function  $g^{-1}$  denotes the inverse of the log link. Significance of  $\delta_{3k}$  will be evaluated with a t-test. Note that model 3 uses the log link as opposed to, for example, the logit link to estimate and test relative risk.

#### 4.11 Evaluation of possible confounded results due to differential co-intervention

The data collected according to the GLORIA protocol are intended to allow a comparison of the effect of prednisolone treatment over placebo in terms of benefit and harm. Given that GLORIA is a pragmatic trial where changes in concomitant treatment (co-interventions for RA, i.e. antirheumatic co-medication) are allowed, an estimation of "pure effects" (i.e. without changes in concomitant treatment) is not possible. When changes in antirheumatic treatment differ between the groups this can result in a confounded estimate of the "pure" effects. Most changes in co-medication can be expected to lower the chance of finding a difference in efficacy between the treatment groups, because negative consequences of being in the placebo group can be countered by changing antirheumatic therapy. For this reason, we also analyze the short-term efficacy of prednisolone in the first three months in a per-protocol population where the chance of confounding is minimized. Note: adverse events leading to stop of study medication are part of the primary harm outcome, and are not covered here.

We will test for potential confounding of the efficacy results. We will not test for confounding of the harm results, because straightforward interpretation is difficult: harm and changes in medication are probably related to each other in a complicated way.

#### 4.11.1 Testing and correcting for differential treatment changes

We plan to check for substantial confounding by comparing the incidence of lasting and substantial changes in co-medication categorized by the reason for change. For practical reasons, we will only consider the first instance of such a change in co-medication. Lasting means we do not consider brief starts or interruptions (i.e., lasting no more than 6 weeks); we also disregard changes in patients stopping the study medication within 3 months following the change.

We will only consider changes that occur in the period starting at 3 months (V2) and 15 months (V6), because the potential for confounding is greatest in this period. Changes before V2 are too early to create confounding, and changes beyond V6 have relatively little effect on the outcome (effect on measurement at V7 and V9). Co-medication includes all disease-modifying antirheumatic drugs (conventional, biologic and targeted), and GC treatment classified as protocol violation and adjudicated in case of oral use.

Oral GC treatment is adjudicated to select occurrences with potential for confounding similar to that of other antirheumatic drugs. Periods of oral treatment up to 3 weeks for RA are equated to one im injection for RA. More than two of either in the period assessed will count as intensification. Oral GC treatment for comorbidity creates less potential for confounding. More than 4 periods of oral treatment for comorbidity lasting no more than 3 weeks will count as intensification. Any period of oral therapy longer than 3 weeks for any indication (RA or otherwise) will also count as intensification.

We distinguish 3 reasons for co-medication changes:

- 1. Lack of efficacy: this includes instances of
  - a. co-medication intensification: increase dose of current antirheumatic drug(s), or adding a new drug (co-medication) to the current treatment, including adjudicated GC treatment classified as protocol violation;
  - b. co-medication switch (replacing one antirheumatic drug with another);
- 2. Adverse event: co-medication switch, or stop of an antirheumatic drug and start of another later; sole dose reduction for adverse event is not considered a substantial change;
- 3. Good efficacy: co-medication taper: decrease dose or stop of current medication(s) without addition of or replacement by another medication.

The remaining patients will be categorized as having no change in co-medication.

For every patient we record and categorize the reason (lack of efficacy, adverse event, good efficacy) for the first change in co-medication in the specified time period. If an adverse event was reported at the moment of change(s) in medication, we will assume that the medication is changed due to adverse events.

Otherwise, if a patient has no reported adverse event(s) at the moment of:

- intensifying or switching the medication: we will assume that the treatment is changed due to lack of efficacy;
- lowering or stopping co-medication: we will assume that the change is due to good efficacy. Situations that are unclear will be adjudicated by the medical monitor before the blind is broken.

The effect of the co-medication change on the expected DAS28 depends on the reason: in case of lack of efficacy or adverse event, the change is expected to lead to a better outcome: a new drug or

an increased dose of the same drug is expected to work better. In case of good efficacy the change is expected to lead to the same or worse outcome: tapering a drug will most likely increase the DAS28 somewhat and may cause a flare.

Therefore, for both treatment groups we will calculate:

- 1. the sum of patients experiencing a co-medication change for lack of efficacy, and for adverse events; and
- 2. the number of patients experiencing a co-medication change for good efficacy.

We will express 1) and 2) as proportion of the total number of patients in each treatment group and compare these between the groups with two Z-tests (each one-sided at p<0.025).

The null hypotheses are:

 $H_{0,4a}$ : The probability of experiencing a co-medication change for lack of efficacy or for adverse events in the placebo group is lower than or equal to the probability in the prednisolone group.  $H_{1,4a}$ : The probability of experiencing a co-medication change for lack of efficacy or for adverse

events in the placebo group is higher than the probability in the prednisolone group.

 $H_{0,4b}$ : The probability of experiencing a co-medication change for good efficacy in the placebo group is higher than or equal to the probability in the prednisolone group.

 $H_{1,4b}$ : The probability of experiencing a co-medication change for good efficacy in the placebo group is lower than the probability in the prednisolone group.

We will assume confounding to the detriment of active treatment if:

- 1.  $H_{0,4a}$  is rejected significantly at p < 0. 025 OR
- 2.  $H_{0,4a}$  is rejected significantly at p < 0.025

Assessing potential for confounding by co-medication changes in the analyses regarding harm of prednisolone is more difficult. Harm and changes in medication are probably related to each other in a complicated way. Therefore, we will not examine this.

#### 4.12 Interpretation rules

The outcomes of benefit (disease activity and damage progression) and harm (number of patients with at least one SAE or other AESI) will be interpreted simultaneously.

The outcomes of benefit will be interpreted as follows (prednisolone group compared to placebo; reference to the specific rejected null hypotheses in parentheses):

- 1. success:
  - a. lower disease activity  $(H_{0,1a})$ AND lower damage score  $(H_{0,2a})$
  - b. lower disease activity OR lower damage score; AND confounding (H<sub>0,4a</sub> or H<sub>0,4b</sub>)
- 2. partial success/tradeoff:
  - a. lower disease activity OR lower damage score AND NO confounding
  - b. NO lower disease AND NO lower damage progression AND confounding
- 3. failure: NO lower disease activity AND NO lower damage score AND NO confounding.

The outcomes of harm will be interpreted as follows:

- 1. success: NO significant increase in AEs
- 2. failure: significant increase in AEs (H<sub>0,3a</sub>)

Combined assessment of benefit and harm

- a. Success: success in benefit and harm
- b. Failure: failure in benefit and harm
- c. Partial success/tradeoff: all other scenarios

For further interpretation of increases in the occurrence of SAE or other AESI in the active treatment group that did not reach significance, we will use the suggestions of the GRADE (Grades of Recommendations, Assessment, Development, and Evaluation) Working Group (Guyatt 2012), upper limit of one-sided 95% confidence interval (CI):

- 1. > 1.3: GC associated with a trend towards greater occurrence;
- 2.  $\leq$  1.2: GC appears to have little effect on the occurrence;
- 3. > 1.2 and  $\le 1.3$ : results failed to demonstrate or exclude a greater occurrence.

In the case of a numerical DECREASE in the occurrence of SAE or other AESI in the active treatment group, a more stringent test for significance will be performed (p<0.025).

For the interpretation of decreases that did not reach significance:

lower limit of one-sided 95% CI:

- 1. < 0.7: GC associated with a trend towards reduced occurrence;
- 2.  $\geq$  0.8: appears to have little effect on the occurrence;
- 3. < 0.8 and  $\ge 0.7$ : results failed to demonstrate or exclude a reduced occurrence.

#### 4.13 Analysis of secondary outcome variables

We will estimate and test for the detrimental effects of prednisolone on bone mass and incident fracture rate.

- 1. Continuous outcomes: bone mass lumbar spine, bone mass hip: analyzed according to model 1
- 2. Discrete outcome: presence of at least one incident compression fracture (by VFA or lateral spine films): analyzed according to model 2

Tests will be one-sided at p<0.05, with Benjamini-Hochberg adjustment for multiple testing.

We will report the results of the other secondary outcome variables descriptively with means/proportions and 95%CI per treatment group per time point.

- 3. Variables measured at every clinic visit
  - a. Continuous outcomes: patient and physician global assessment of disease activity, joint counts (swollen joints and tender joints), acute phase reactants (C-reactive protein (CRP) and erythrocyte sedimentation rate (ESR)); vital signs, lab (blood) variables; adherence by pill count and by electronic adherence cap.
  - b. Discrete outcomes: patients with at least one instance of remission; of minimal disease activity; patients with at least one long-term period (2 consecutive instances 6 months apart) of remission; of minimal disease activity
- 4. Variables measured at every visit (clinic and remote):
  - a. Continuous outcomes: severity and duration of morning stiffness, RA Impact of disease (total score, and components pain and fatigue analyzed separately), RAPID3 index, EuroQoL, m(HAQ)
  - b. Discrete outcomes: discontinuations of study drug, of with reason; all changes of antirheumatic treatment, with reason; joint replacement surgery
  - c. Expressed as survival curve: discontinuation of study drug over time
- 5. Variables measured at baseline and end of study:
  - a. Continuous outcomes: DAS44, SF36 (domains and summary mental and physical component scores), 57-symptom list;
  - b. Discrete outcome: number of incident compression fractures (by VFA or lateral spine films)
- 6. Variables measured only at baseline:
  - a. Continuous/discrete:
    - Demographics, education and medical history; Morisky medication adherence scale (MMAS-8), health literacy, arthritis helplessness index questionnaires; number of prevalent vertebral fractures (by VFA or lateral spine films), distribution of % height loss in vertebrae with fractures.
- 7. Response indices calculated at 3 months in the PP analysis (discrete): ACR20, 50, 70; EULAR response.

#### 5 Interim analyses

No interim analyses were planned. However, we performed a new sample size calculation based on blinded AE incidence rates halfway through the trial (see below).

#### 6 Sample size and power calculations

In the main GLORIA trial, 225 patients per treatment group will be entered (total 450 patients).

In the chosen analysis strategy (see section 4), to detect differences in benefit (disease activity, radiographs) extensive RA trial experience (both for GC and other agents) has shown a sample size of 200 patients per group is amply sufficient. For example, in the CAPRA-2 study that compared modified release prednisone 5mg/d against placebo, the prednisone group had 231 patients, the placebo group 119 patients. The change in DAS28 after 3 months of treatment was –1.15 in the prednisone group, –0.63 in the placebo group; difference –0.52 (SE 0.13, p<0.001) (Buttgereit, 2013). However, the true incidence of adverse events (AEs) for GCs is currently unknown. Most relevant data to assess sample size adequacy for this study come from the reported CAMERA-2 trial (Bakker, 2012). This trial randomized 236 early RA patients to tight-control high-dose methotrexate plus 10 mg prednisolone or placebo for two years. Interestingly, 22% of placebo patients compared to only 14% of prednisolone patients reported at least one serious AE or clinical event as defined in our protocol.

The original protocol used a base case expectation for a total of 20% of patients experiencing at least one event over two years in the placebo group and calculated a need for 400 patients in each treatment group, to have about 80% power to detect an increase of 7% (from 20% to 27% events; 90% power for an increase of 9%). However, based on our current experience the sample can be decreased to about 450 instead of 800.

#### Elaboration:

In December 2018 we had >400 patients in the trial with a mean follow up of 9 months, and we had 84 cases with at least one serious adverse event or an event of special interest (the primary harm outcome). A simple extrapolation leads to an estimated rate of about 49% over 2 years (pooled over the whole blinded trial population, i.e. both treatment groups taken together). We have also performed life table analysis, which accounts for patients stopping prematurely; this analysis leads to an estimated rate of 40% (95% confidence interval: 30%-50%).

Given the above we can now assume with confidence that the base rate of patients with events in the placebo group will be substantially higher than originally predicted. This adds power to the trial: we need only between 400 and 450 patients to detect the originally targeted contrast of 27.5%/20%= relative risk of 1.38 (Table 1). At the expected pooled event rate of 40%, with 400 patients we have 80% power to detect a difference of 12% between placebo and prednisolone: i.e. placebo 34% and prednisolone 46%, a relative risk of 1.35. The results are better with 450 patients, and when the event rate is higher (Table 1). At the moment of submission of the amendment trial recruitment has been closed on December 31, 2018 at a total of 452 patients.

Table 1. Sample size scenarios (one-sided alpha 5%).

| expected event ra | ate over 2 years | | | | |
|---|---|---|---|---|---|
| (% unique | patients | | with power 80%, | | |
| with at least | one event) | detectable rate | n predn group | Relativ | e Risk |
| pooled | placebo | n=400 | n=450 | n=400 | n=450 |
| 30% | 26% | 38% | 37% | 1,47 | 1,43 |
| 35% | 30% | 42% | 41% | 1,40 | 1,37 |
| 40% | 34% | 46% | 45% | 1,35 | 1,32 |
| 45% | 39% | 52% | 52% | 1,31 | 1,31 |
| 50% | 43% | 55% | 55% | 1,28 | 1,28 |

## 7 Tables, listings and figures

Below are the titles for the planned study tables, figures, and listings.

| Table 1 | Patient distribution |
|---|---|
| Table 2.A | Patient distribution by center (ITT) |
| Table 2.B | Patient distribution by center (PP) |
| Table 3.A | Demographics and baseline characteristics (ITT) |
| Table 3.B | Demographics and baseline characteristics (PP) |
| Table 4 | Health literacy |
| Table 5 | Morisky medication adherence scale (MMAS-8) |
| Table 6 | Arthritis helplessness index Table 7 .A Medical history (ITT) |
| Table 7.B | Medical history (PP) |
| Table 8.A | DAS28 scores (ITT) |
| Table 8.B | DAS28 scores (PP) |
| Table 9 | Mixed effects model of time-averaged DAS28 (ITT) |
| Table 10 | DAS44 scores (ITT)Table 11.A Swollen joints 28 joint count (ITT) |
| Table 11.B | Swollen joints 28 joint count (PP) |
| Table 12.A | Tender joints 28 joint count (ITT) |
| Table 12.B | Tender joints 28 joint count (PP) |
| Table 13.A | Patient global assessment of disease activity (ITT) |
| Table 13.B | Patient global assessment of disease activity (PP) |
| Table 14.A | Physician global assessment of disease activity (ITT) |
| Table 14.B | Physician global assessment of disease activity (PP) |
| Table 15.A | CRP (ITT) |
| Table 15.B | CRP (PP) |
| Table 16.A | ESR (ITT) |
| Table 16.B | ESR (PP)Table 17 EULAR response (PP) |
| Table 18 | ACR response (PP) |
| Table 19.A | Minimal disease activity (ITT) |
| Table 19.B | Minimal disease activity (PP) |
| Table 20 | Total Sharp/van der Heijde damage score of hands and forefeet radiographs (ITT) |
| Table 21 | Morning stiffness (ITT) |
| Table 22 | SF-36 questionnaire (ITT) |
| Table 23 | RAID questionnaire (ITT) |
| Table 24 | (Modified) Health Assessment Questionnaire ((m)HAQ) (ITT) |
| Table 25 | RAPID3 (ITT) |
| Table 26 | EuroQoL questionnaire (ITT) |
| Table 27 | 57-symptom list (ITT) |
| Table 28.A | Laboratory results in SI and original units (ITT) |
| Table 28.B | Laboratory results in SI and original units (SAF) |
| Table 29.A | Vital signs (ITT) |
| Table 29.B | Vital signs (SAF) |
| Table 30.A | Adherence (ITT) |
| Table 30.B | Adherence (PP) |

| Table 30.C | Adherence (SAF) |
|---|---|
| Table 31 | Concomitant medications summary (ITT) |
| Table 32 | Bone mass (ITT) |
| Table 33 | Number of prevalent vertebral fractures (by VFA or lateral spine films) (ITT) |
| Table 34 | Distribution of % height loss in vertebrae with fractures |
| Table 35 | Joint replacement surgery (ITT) |
| Table 36.A | AEs, SAEs and other AEs of special interest summary (ITT) |
| Table 36.B | AEs, SAEs and other AEs of special interest summary (SAF) |
| Table 36.C | AEs, SAEs and other AEs of special interest (ITT) |
| Table 36.D | AEs, SAEs and other AEs of special interest (SAF) |
| Table 37 | Presence of SAE or other AE of special interest (ITT) |

| Table title | Number | Population | Endpoint | Time points or | Covariates or | Type of variable | Summary |
|---|---|---|---|---|---|---|---|
| | | | | how to conglomerate | subgroups | | statistics |
| Patient distribution | 1 | Intent-to-treat population | Distribution | Baseline | - | Dichotomous | % (n) |
| Patient | 2A | Intent-to-treat | Distribution | Baseline | Treatment group | Dichotomous | % (n) |
| distribution by center | | population | | | | | |
| Patient | 2B | Per-protocol | Distribution | Baseline | Treatment group | Dichotomous | % (n) |
| distribution by center | | population | | | | | |
| Demographics and baseline | 3A + 3B | 3A. Intent-to-<br>treat | Age | Baseline | Treatment group | Continuous | Mean (SD)<br>(median, min, |
| characteristics | | population<br>3B. Per- | | | | | max if data are<br>non-normal |
| | | protocol | | | | | distributed), n |
| | | | Sex | Baseline | Treatment group | Dichotomous | % (n) female |
| | | | Smoking status | Baseline | Treatment group | Categorical | Current: % (n)<br>Previous: % (n)<br>Never: % (n) |

| Table title | Number | Population | Endpoint | Time points or how to conglomerate | Covariates or subgroups | Type of variable | Summary statistics |
|---|---|---|---|---|---|---|---|
| | | | Alcohol intake (units per week) | Baseline | Treatment group | Categorical | Every day: % (n) 5-6 days per |
| | | | | | | | week: % (n) |
| | | | | | | | week: % (n) |
| | | | | | | | 1-2 days per |
| | | | | | | | week: % (n) |
| | | | | | | | 1-3 days per |
| | | | | | | | /1 day per |
| | | | | | | | month: % (n) |
| | | | | | | | Nevel . 70 (II) |
| | | | Possession of smartphone | Baseline | Treatment group | Dichotomous | % (n) |
| | | | Education level | Baseline | Treatment group | Categorical | % (n) higher education |
| | | | Duration of | Baseline | Treatment group | Continuous | Mean (SD) |
| | | | rheumatoid arthritis<br>(months) | | | | (median, min, |
| | | | | | | | non-normal |
| | | | | | | | distributed), fi |
| | | | Rheumatoid factor<br>status | Baseline | Treatment group | Dichotomous | % (n), positive |
| | | | Anti-CCP status | Baseline | Treatment group | Dichotomous | % (n), positive |

| Table title | Number | Population | Endpoint | Time points or | Covariates or | Type of variable | Summary |
|---|---|---|---|---|---|---|---|
| | | | | how to conglomerate | subgroups | | statistics |
| | | | Evidence of structural | Baseline | Treatment group | Categorical | % (n), yes |
| | | | joint damage | | | | |
| | | | Previous related surgical procedures | Baseline | Treatment group | Categorical | % (n), yes |
| | | | surgical procedures | | | | |
| | | | Previous | Baseline | Treatment group | Dichotomous | % (n), yes |
| | | | glucocorticoid<br>treatment | | | | |
| | | | Previous NSAID | Baseline | Treatment group | Dichotomous | % (n), yes |
| | | | creatilient | | | | |
| | | | Previous DMARD treatment | Baseline | Treatment group | Dichotomous | % (n), yes |
| | | | Previous biological | Baseline | Treatment group | Dichotomous | % (n), yes |
| | | | treatment | | | | |
| | | | Number of | Baseline | Treatment group | Continuous | Mean (SD) |
| | | | comorbidities | | | | (median, min, |
| | | | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |
| | | | DAS28 | Baseline | Treatment group | Continuous | Mean (SD) |
| | | | | | | | (median, min, |
| | | | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |

| distributed), n | | | | | | | |
|---|---|---|---|---|---|---|---|
| non-normal | | | | | | | |
| max if data are | | | | | | | |
| (median, min, | | | | severity | | | |
| Mean (SD) | Continuous | Treatment group | Baseline | Morning stiffness | | | |
| distributed) | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | | | | |
| (median, min, | | | | duration in minutes | | | |
| Mean (SD) | Continuous | Treatment group | Baseline | Morning stiffness, | | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | | | | |
| (median, min, | | | | | | | |
| Mean (SD) | Continuous | Treatment group | Baseline | CRP | | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | | | | |
| (median, min, | | | | | | | |
| Mean (SD) | Continuous | Treatment group | Baseline | ESR | | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | | | | |
| (median, min, | | | | | | | |
| Mean (SD) | Continuous | Treatment group | Baseline | Swollen joint count | | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | | | | |
| (median, min, | | | | | | | |
| Mean (SD) | Continuous | Treatment group | Baseline | Tender joint count | | | |
| Statistics | | 342810473 | conglomerate | | | | |
| statistics | | cubarounc | bow +0 | 1 | - | | |
| Summary | Type of variable | Covariates or | Time points or | Endpoint | Population | Number | Table title |

| distributed), n | | | | | | | |
|---|---|---|---|---|---|---|---|
| non-normal | | | | | | | |
| max if data are | | | | | | | |
| (median, min, | | | | | | | |
| Mean (SD) | Continuous | Treatment group | Baseline | EQ-5D | | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | | | | |
| (median, min, | | | | | | | |
| Mean (SD) | Continuous | Treatment group | Baseline | RAID | | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | | | | |
| (median, min, | | | | | | | |
| Mean (SD) | Continuous | Treatment group | Baseline | HAQ (scale 0-3) | | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | | | | |
| (median, min, | | | | | | | |
| Mean (SD) | Continuous | Treatment group | Baseline | Pain (scale 0-10) | | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | activity (scale 0-10) | | | |
| (median, min, | | | | assessment of disease | | | |
| Mean (SD) | Continuous | Treatment group | Baseline | Physician global | | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | activity (scale 0-10) | | | |
| (median, min, | | | | assessment of disease | | | |
| Mean (SD) | Continuous | Treatment group | Baseline | Patient global | | | |
| SIGUSTICS | | subgroups | conglomerate | | | | |
| otatiotics , | 7000 | cubarruna ci | b) | : | | | |
| Silmmary | Type of variable | Covariates or | Time points or | Endpoint . | Population | Number | Tahle title |

| Table title | Niimhar | Donulation | Endpoint | Time points or | Covariates or | Type of variable | Simmary |
|---|---|---|---|---|---|---|---|
| | 3 | | | how to | subgroups | . The containing | statistics |
| | | | | Coligioniciate | | | |
| | | | SF36 | Baseline | Treatment group | Continuous | Mean (SD) |
| | | | | | | | (median, min, |
| | | | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |
| Health literacy | 4 | Intent-to-treat | Health literacy | Baseline | Treatment group | Continuous | Mean (SD) |
| | | population | | | | | (median, min, |
| | | | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |
| Morisky | Л | Intent-to-treat | Morisky medication | Baseline | Treatment group | Continuous | Mean (SD) |
| medication | | population | adherence scale | | | | (median, min, |
| adherence scale | | | | | | | max if data are |
| (MMAS-8) | | | | | | | non-normal |
| | | | | | | | distributed), n |
| Arthritis | 6 | Intent-to-treat | Arthritis helplessness | Baseline | Treatment group | Categorical | -Low: % (n) |
| helplessness | | population | index | | | | -Normal: % (n) |
| index | | | | | | | -High: % (n) |
| Medical history | 7A | Intent-to-treat | Number of | Baseline | Treatment group | Continuous | % (n) |
| | | population | comorbidities per | | | | |
| | | | organ system class | | | | |
| | | | Top 3 of most | Baseline | | | 1. % (n) |
| | | | common comorbidity | | | | 2. % (n) |
| | | | categories | | | | 3. % (n) |
| | 7B | Per-protocol | Number of | Baseline | Treatment group | Continuous | % (n) |
| | | population | comorbidities per | | | | |
| | | | organ system class | | | | |
| Table title | Number | Population | Endpoint | Time points or | Covariates or | Type of variable | Ynemmus |
|---|---|---|---|---|---|---|---|
| | | | | how to | subgroups | | statistics |
| | | | | conglomerate | | | |
| | | | Top 3 of most | Baseline | Treatment group | Continuous | 1. % (n) |
| | | | common comorbidity | | | | 2. % (n) |
| | | | categories | | | | 3. % (n) |
| DAS28 scores | 8A | Intent-to-treat | DAS28 score | 0, 3, 6, 12, 18, | Treatment group | Continuous | Mean (SD) |
| | | population | | 24 months | | | (median, min, |
| | | | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |
| | | | Change in DAS28 score | 0-3 months | Treatment group | Continuous | Mean (SD) |
| | | | | | | | (median, min, |
| | | | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |
| | | | Change in DAS28 score | 0-24 months | Treatment group | Continuous | Mean (SD) |
| | | | | | | | (median, min, |
| | | | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |
| | 8B | Per-protocol | DAS28 score | 0, 3 months | Treatment group | Continuous | Mean (SD) |
| | | population | | | | | (median, min, |
| | | | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |
| | | | Change in DAS28 score | 0-3 months | Treatment group | Continuous | Mean (SD) |
| | | | | | | | (median, min, |
| | | | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |

| Table title | Number | Population | Endpoint | Time points or | Covariates or | Type of variable | Summary |
|---|---|---|---|---|---|---|---|
| | | | | how to | subgroups | | statistics |
| | | | | conglomerate | | | |
| Mixed effects | 9 | Intent-to-treat | DAS28 score | 0, 3, 6, 9, 12, | Treatment group | Continuous | Value, |
| model of time- | | population | | 18, 24 months | | | Standard |
| averaged DAS28 | | | | | | | Error, Df, p- |
| | | | | | | | value |
| DAS44 scores | 10 | Intent-to-treat | DAS44 score | 0 months | Treatment group | Continuous | Mean (SD) |
| | | population | | | | | (median, min, |
| | | | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |
| | | Intent-to-treat | Change in DAS44 score | 0-24 months | Treatment group | Continuous | Mean (SD) |
| | | population | | | | | (median, min, |
| | | | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |
| Swollen joints 28 | 11A | Intent-to-treat | Number of swollen | 0, 3, 6, 9, 12, | Treatment group | Continuous | Mean (S |
| joint count | | population | joints | 18, 24 months | | | 95% CI |
| | | | | | | | (median, min, |
| | | | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |
| | 11B | Per-protocol | Number of swollen | 0, 3 months | Treatment group | Continuous | Mean ( |
| | | population | joints | | | | 95% CI |
| | | | | | | | (median, min, |
| | | | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |

| Table title | Number | Population | Endpoint | Time points or how to conglomerate | Covariates or subgroups | Type of variable | Summary statistics |
|---|---|---|---|---|---|---|---|
| Tender joints 28 joint count | 12A | Intent-to-treat population | Number of tender joints | 0, 3, 6, 9, 12,<br>18, 24 months | Treatment group | Continuous | Mean (SD) +<br>95% Cl |
| | | | | | | | (median, min,<br>max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |
| | 12B | Per-protocol | Number of tender | 0, 3 months | Treatment group | Continuous | Mean (SD) + |
| | | population | joints | | | | 95% CI |
| | | | | | | | (median, min, |
| | | | | | | | max if data are |
| | | | | | | | non-normal |
| Patient global | 13A | Intent-to-treat | Patient global | 0, 3, 6, 9, 12, | Treatment group | Continuous | Mean (SD) + |
| assessment of | | population | assessment of disease | 18, 24 months | | | 95% CI |
| disease activity | | | activity | | | | (median, min, |
| | | | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |
| | 13B | Per-protocol | Patient global | 0, 3 months | Treatment group | Continuous | Mean (SD) + |
| | | population | assessment of disease | | | | 95% CI |
| | | | activity | | | | (median, min, |
| | | | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | מוסנווסמנכמ/, וו |
| Physician global assessment of | 14A | Intent-to-treat | Physician global assessment of disease | 0, 3, 6, 9, 12,<br>18, 24 months | Treatment group | Continuous | 95% CI |
| disease activity | | | activity | | | | (median, min, |
| | | | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |

| Table title | Number | Population | Endpoint | Time points or | Covariates or | Type of variable | Summary |
|---|---|---|---|---|---|---|---|
| | | • | - | how to conglomerate | subgroups | : | statistics |
| | 14B | Per-protocol population | Physician global assessment of disease | 0, 3 months | Treatment group | Continuous | Mean (SD) +<br>95% Cl |
| | | | activity | | | | (median, min, |
| | | | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |
| CRP | 15A | Intent-to-treat | CRP | 0, 3, 6, 9, 12, | Treatment group | Continuous | Mean (SD) + |
| | | population | | 18, 24 months | | | 95% CI |
| | 15B | Per-protocol | CRP | 0, 3 months | Treatment group | Continuous | (median, min, |
| | | population | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |
| ESR | 16A | Intent-to-treat | ESR | 0, 3, 6, 9, 12, | Treatment group | Continuous | Mean (SD) + |
| | | population | | 18, 24 months | | | 95% CI |
| | 16B | Per-protocol | ESR | 0, 3 months | Treatment group | Continuous | (median, min, |
| | | population | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |
| EULAR response | 17 | Per-protocol | EULAR response | 3 months | Treatment group | Categorical | Good: % (n) |
| | | population | | | | | Moderate: % |
| | | | | | | | (n) |
| | | | | | | | None: % (n) |
| American College | 18 | Per-protocol | ACR20 response | 3 months | Treatment group | Dichotomous | % (n), yes |
| of Rheumatology | | population | | | | | |
| (ACR) response | | | | | | | |
| | | | ACR50 response | 3 months | Treatment group | Dichotomous | % (n), yes |
| | | | ACR70 response | 3 months | Treatment group | Dichotomous | % (n), yes |
| Minimal disease | 19A | Intent-to-treat | Minimal disease | 3, 6, 12, 18, | Treatment group | Dichotomous | % (n), yes |
| activity | | population | activity | 24months | | | |

| nerate<br>, 18, 24<br>24<br>24<br>; 18,<br>ths<br>hs<br>onths | Table title | Number | Population | Endpoint | Time points or | Covariates or | Type of variable | Summary |
|---|---|---|---|---|---|---|---|---|
| Boolean remission 3, 6, 12, 18, 24 Treatment group characteristics and the pisode months and the pisode months and the pisode months activity 3, 6, 12, 18, 24 Treatment group activity 3, 6, 12, 18, 24 Treatment group hadron activity 3, 6, 12, 18, 24 Treatment group activity 3, 6, 12, 18, 24 Treatment group activity 3, 6, 12, 18, 24 Treatment group activity 3 months Treatment group population activity 3 months Treatment group lands (SDAI) Mitent-to-treat Sharp/van der Heijde 0, 24 months Treatment group population der Heijde damage score der Heijde damage score activity 3 months Treatment group population der Heijde damage score der Heijde damage score activity 3 months Treatment group der Heijde damage score activity 3 months Treatment group der Heijde damage score activity 3 months Treatment group der Heijde damage score activity 3 months Treatment group der Heijde damage score activity 3 months Treatment group activity 3 months Treatment group der Heijde damage score activity 3 months Treatment group activity 3 months Treatment group activity 3 months 3 months Treatment group activity 3 months 3 months 4 months 4 months 4 months 5 months 5 months 5 months 5 months 6 months 6 months 7 months 7 meatment group 8 months 7 months 7 meatment group 9 months | | | | | how to conglomerate | subgroups | | statistics |
| episode Long-term Boolean L2, 18, 24 Treatment group Index (SDAI) 198 Per-protocol Minimal disease 199 Population Boolean remission Boo | | | | Boolean remission | 3, 6, 12, 18, 24 | Treatment group | Dichotomous | % (n), yes |
| Long-term Boolean 12, 18, 24 Treatment group months Simple Disease Activity 3, 6, 12, 18, Treatment group 24months 19B Per-protocol Minimal disease 3 months Treatment group 24months Simple Disease Activity 3 months Treatment group 24months Simple Disease Activity 3 months Treatment group 25mple Disease Activity 3 months 25mple Disease Act | | | | episode | months | | | |
| remission months Simple Disease Activity 3,6,12,18, Treatment group 24months | | | | Long-term Boolean | 12, 18, 24 | Treatment group | Dichotomous | % (n), yes |
| Simple Disease Activity 3, 6, 12, 18, Treatment group nindex (SDAI) 24months 19B Per-protocol Minimal disease 3 months Treatment group population activity 9,000 activity 24months Treatment group episode 15mple Disease Activity 3 months Treatment group nindex (SDAI) 3 months Treatment group population damage score 15mplyvan der Heijde 0,24 months Treatment group der Heijde damage score 15mplyvan 0-24 months Treatment group der Heijde damage score 15,18,21,24 months 15mplyvan 0-3,6,9,12, 15,18,21,24 months 15mplyvan 0,3,6,9,12, 15,18,21,24 months 15mplyvan 15,18,21,24 months 15mplyvan 15,18,21,24 months 15mplyvan 15mplyvan 15,18,21,24 months 15mplyvan 15mplyv | | | | remission | months | | | |
| 19B Per-protocol Minimal disease 3 months Treatment group population activity 3 months Treatment group episode Simple Disease Activity 3 months Treatment group Index (SDAI) 19B Per-protocol Minimal disease 3 months Treatment group episode Simple Disease Activity 3 months Treatment group Index (SDAI) 19B Per-protocol Minimal disease Activity 3 months Treatment group Index (SDAI) 19B Per-protoco | | | | Simple Disease Activity | 3, 6, 12, 18, | Treatment group | Dichotomous | % (n), yes |
| 19B Per-protocol Minimal disease 3 months Treatment group population activity Boolean remission 3 months Treatment group episode Simple Disease Activity 3 months Treatment group Index (SDAI) 3 months Treatment group 4 months Treatment group 5 more of Change in Sharp/van der Heijde damage score Change in Sharp/van 0-24 months Treatment group 6 morning stiffness 21 Intent-to-treat Duration (minutes) of population 0, 3, 6, 9, 12, months months Treatment group 15, 18, 21, 24 months months Treatment group 15, 18, 21, 24 months months Treatment group 15, 18, 21, 24 months months Treatment group 15, 18, 21, 24 months | | | | Index (SDAI) | 24months | | | |
| population activity Boolean remission 3 months Treatment group episode Simple Disease Activity 3 months Treatment group Index (SDAI) Syvan 20 Intent-to-treat Sharp/van der Heijde 0, 24 months Treatment group population damage score Change in Sharp/van 0-24 months Treatment group der Heijde damage score Intent-to-treat Duration (minutes) of population morning stiffness 21 Intent-to-treat population morning stiffness 21 population morning stiffness 21 morning stiffness 21 population morning stiffness 21 morning stiffness Intents proup months months | | 19B | Per-protocol | Minimal disease | 3 months | Treatment group | Dichotomous | % (n), yes |
| Boolean remission episode Simple Disease Activity 3 months Treatment group Index (SDAI) J/van 20 Intent-to-treat Sharp/van der Heijde 0, 24 months Treatment group damage score Secore Change in Sharp/van 0-24 months Treatment group der Heijde damage score Intent-to-treat Duration (minutes) of population morning stiffness 21 Intent-to-treat population morning stiffness months months Treatment group 15, 18, 21, 24 months morning stiffness months | | | population | activity | | | | |
| episode Simple Disease Activity 3 months Index (SDAI) J/van 20 Intent-to-treat Sharp/van der Heijde o, 24 months Treatment group on the population damage score Change in Sharp/van o-24 months Change in Sharp/van o-24 months Ger Heijde damage score Intent-to-treat population morning stiffness Intent-to-treat population morning stiffness months Treatment group on the population on the population morning stiffness months | | | | Boolean remission | 3 months | Treatment group | Dichotomous | % (n), yes |
| Simple Disease Activity 3 months Treatment group Index (SDAI) 15 Change in Sharp/van der Heijde damage score Change in Sharp/van der Heijde damage score O-24 months Treatment group 15 Change in Sharp/van der Heijde damage score Duration (minutes) of population | | | | episode | | | | |
| J/van 20 Intent-to-treat Sharp/van der Heijde O, 24 months Treatment group population damage score ore of Change in Sharp/van O-24 months Treatment group der Heijde damage score Iiffness 21 Intent-to-treat population morning stiffness morning stiffness morning stiffness morning stiffness morning stiffness months | | | | Simple Disease Activity | 3 months | Treatment group | Dichotomous | % (n), yes |
| ore of core | | | | Index (SDAI) | | | | |
| ore of Change in Sharp/van 0-24 months Treatment group der Heijde damage score | Total Sharp/van | 20 | Intent-to-treat | Sharp/van der Heijde | 0, 24 months | Treatment group | Continuous | Mean (SD) + |
| Change in Sharp/van 0-24 months Treatment group der Heijde damage score 21 Intent-to-treat population morning stiffness months Change in Sharp/van 0-24 months Treatment group 0-3, 6, 9, 12, Treatment group months | der Heijde | | population | damage score | | | | 95% CI |
| Change in Sharp/van 0-24 months Treatment group der Heijde damage score 21 Intent-to-treat population morning stiffness months months months | damage score of | | | | | | | (median, min, |
| Change in Sharp/van 0-24 months Treatment group der Heijde damage score 21 Intent-to-treat population morning stiffness population morning stiffness months | hands and | | | | | | | max if data are |
| Change in Sharp/van der Heijde damage score 21 Intent-to-treat population morning stiffness population Change in Sharp/van 0-24 months Treatment group 0,3,6,9,12, 15,18,21,24 months | forefeet | | | | | | | non-normal |
| Change in Sharp/van 0-24 months Treatment group der Heijde damage score 21 Intent-to-treat population morning stiffness months months months | radiographs | | | | | | | distributed), n |
| der Heijde damage score 21 Intent-to-treat population morning stiffness mornths der Heijde damage score 0, 3, 6, 9, 12, Treatment group months | | | | Change in Sharp/van | 0-24 months | Treatment group | Continuous | Mean (SD) + |
| 21 Intent-to-treat population morning stiffness population morning stiffness months | | | | der Heijde damage | | | | 95% CI |
| 21 Intent-to-treat Duration (minutes) of 0, 3, 6, 9, 12, population morning stiffness 15, 18, 21, 24 months | | | | score | | | | (median, min, |
| 21 Intent-to-treat Duration (minutes) of 0, 3, 6, 9, 12, population morning stiffness months | | | | | | | | max if data are |
| 21 Intent-to-treat Duration (minutes) of 0, 3, 6, 9, 12, population morning stiffness months | | | | | | | | non-normal |
| 21 Intent-to-treat Duration (minutes) of population morning stiffness months 15, 18, 21, 24 months | | | | | | | | distributed), n |
| population morning stiffness 15, 18, 21, 24 months | Morning stiffness | 21 | Intent-to-treat | Duration (minutes) of | 0, 3, 6, 9, 12, | Treatment group | Continuous | + (SD) + |
| | | | population | morning stiffness | 15, 18, 21, 24 | | | 95% CI |
| | | | | | months | | | (median, min, |
| | | | | | | | | max if data are |
| | | | | | | | | non-normal |
| | | | | | | | | distributed), n |

| Table title | Number | Population | Endpoint | Time points or | Covariates or | Type of variable | Summary |
|---|---|---|---|---|---|---|---|
| | | - | | how to conglomerate | subgroups | : | statistics |
| | | Intent-to-treat | Severity of morning | 0, 3, 6, 9, 12, | Treatment group | Continuous | Mean (SD) + |
| | | population | | 15, 18, 21, 24 | | | 95% CI |
| | | | | months | | | (median, min, |
| | | | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |
| SF-36 | 22 | Intent-to-treat | SF-36 physical | 0 months | Treatment group | Continuous | Mean (SD) + |
| | | population | functioning score | | | | 95% CI |
| | | | | | | | (median, min, |
| | | | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |
| | | Intent-to-treat | Change in SF-36 | 0-24 months | Treatment group | Continuous | Mean (SD) + |
| | | population | physical functioning | | | | 95% CI |
| | | | score | | | | (median, min, |
| | | | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |
| | | Intent-to-treat | SF-36 role-physical | 0 months | Treatment group | Continuous | Mean (SD) |
| | | population | score | | | | (median, min, |
| | | | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |
| | | Intent-to-treat | Change in SF-36 role- | 0-24 months | Treatment group | Continuous | Mean (SD) |
| | | population | physical score | | | | (median, min, |
| | | | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |

| 200 | | | | | | | |
|---|---|---|---|---|---|---|---|
| max if data are | | | | | | | |
| (median, min, | | | | vitality score | population | | |
| Mean (SD) | Continuous | Treatment group | 0-24 months | Change in SF-36 | Intent-to-treat | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | | | | |
| (median, min, | | | | | population | | |
| Mean (SD) | Continuous | Treatment group | 0 months | SF-36 vitality score | Intent-to-treat | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | | | | |
| (median, min, | | | | general health score | population | | |
| Mean (SD) | Continuous | Treatment group | 0-24 months | Change in SF-36 | Intent-to-treat | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | | | | |
| (median, min, | | | | score | population | | |
| Mean (SD) | Continuous | Treatment group | 0 months | SF-36 general health | Intent-to-treat | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | | | | |
| (median, min, | | | | pain score | population | | |
| Mean (SD) | Continuous | Treatment group | 0-24 months | Change in SF-36 bodily | Intent-to-treat | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | | | | |
| (median, min, | | | | score | population | | |
| Mean (SD) | Continuous | Treatment group | 0 months | SF-36 bodily pain | Intent-to-treat | | |
| | | 0 - 1 | conglomerate | | | | |
| statistics | : | subgroups | how to | | | | |
| Summary | Type of variable | Covariates or | Time points or | Endpoint | Population | Number | Table title |

| max if data are | | | | | | | |
|---|---|---|---|---|---|---|---|
| (median, min, | | | | mental health score | population | | |
| Mean (SD) | Continuous | Treatment group | 0-24 months | Change in SF-36 | Intent-to-treat | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | | | | |
| (median, min, | | | | score | population | | |
| Mean (SD) | Continuous | Treatment group | 0 months | SF-36 mental health | Intent-to-treat | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | | | | |
| (median, min, | | | | emotional score | population | | |
| Mean (SD) | Continuous | Treatment group | 0-24 months | Change in SF-36 role- | Intent-to-treat | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | | | | |
| (median, min, | | | | score | population | | |
| Mean (SD) | Continuous | Treatment group | 0 months | SF-36 role-emotional | Intent-to-treat | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | | | | |
| (median, min, | | | | functioning score | population | | |
| Mean (SD) | Continuous | Treatment group | 0-24 months | Change in SF-36 social | Intent-to-treat | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | | | | |
| (median, min, | | | | functioning score | population | | |
| Mean (SD) | Continuous | Treatment group | 0 months | SF-36 social | Intent-to-treat | | |
| | | 0.000 | conglomerate | | | | |
| statistics | : | subgroups | how to | | • | | |
| Summary | Type of variable | Covariates or | Time points or | Endpoint | Population | Number | Table title |

| طان الحال العالم | | | | | | | |
|---|---|---|---|---|---|---|---|
| non-normal | | | | | | | |
| (median, min, | | | 24months | | | | |
| 95% CI | | | 15, 18, 21, | | population | | |
| Mean (SD) + | Continuous | Treatment group | 0, 3, 6, 9, 12, | RAID total score | Intent-to-treat | 23 | RAID |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | summary score | | | |
| (median, min, | | | | mental component | population | | |
| Mean (SD | Continuous | Treatment group | 0-24 months | Change in SF-36 | Intent-to-treat | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | score | | | |
| (median, min, | | | | component summary | population | | |
| Mean (SD) | Continuous | Treatment group | 0 months | SF-36 mental | Intent-to-treat | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | summary score | | | |
| (median, | | | | physical component | population | | |
| Mean (SD) | Continuous | Treatment group | 0-24 months | Change in SF-36 | Intent-to-treat | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | score | | | |
| (median, min, | | | | component summary | population | | |
| Mean (SD) | Continuous | Treatment group | 0 months | SF-36 physical | Intent-to-treat | | |
| | | | conglomerate | | | | |
| statistics | | subgroups | how to | | | | |
| Summary | Type of variable | Covariates or | lime points or | Endpoint | Population | Number | Table title |

| RAID pain score RAID pain score 15.18. 21. 24 months 24 intent-to-treat population 25 intent-to-treat population 26 intent-to-treat population 27 population 28 population 29 population 29 population 20 population 20 point pain score population 20 paintent score population 20 paintent score population 21 population 22 population 23 population 24 population 25 population 26 paintent group population 27 preatment group population 28 population 29 population 20 population 20 population 20 population 21 population 22 paintent group population 23 population 24 population 25 population 26 population 27 preatment group population 28 population 29 population 20 population 20 population 20 population 20 population 21 population 30 population 31 population 42 population 43 population 44 population 45 population 45 population 46 population 47 population 57 population 58 population 59 population 60 | Table title | Number | Population | Endpoint | Time points or | Covariates or | Type of variable | vaemmis |
|---|---|---|---|---|---|---|---|---|
| RAID pain score 0, 3, 6, 9, 12, 24 Intent-to-treat population 25 Intent-to-treat population 26 Intent-to-treat population 27 Intent-to-treat population 28 Intent-to-treat population 29 Intent-to-treat population 20 Intent-to-treat population 20 Intent-to-treat population 21 Intent-to-treat population 22 Intent-to-treat population 23 Intent-to-treat population 24 Intent-to-treat population 25 Intent-to-treat population 26 Intent-to-treat population 27 Intent-to-treat population 28 Intent-to-treat population 29 Intent-to-treat population 10 J. 18, 21, 24 Intent group population 15 J. 18, 21, 24 Intent group population 26 Intent-to-treat population 27 Intentment group population 28 Intent-to-treat population 19 J. 18 J. 19 J. 24 Intentment group population 19 J. 18 J. 21 J. 3 J. 3 J. 3 J. 3 J. 3 J. 3 J. 3 J. | | | - | - | how to conglomerate | subgroups | | statistics |
| 24 Intent-to-treat population PAPID3 index score population Population Popula | | | | RAID pain score | 0, 3, 6, 9, 12, | Treatment group | Continuous | Mean (SD) + |
| 24 Intent-to-treat population PAPID3 index score population Population Popula | | | | | 15, 18, 21, | | | 95% CI |
| RAID fatigue score 0, 3, 6, 9, 12. Treatment group Continuous 15, 18, 21, 24 Intent-to-treat population population 25 Intent-to-treat Population Population 26 Intent-to-treat population 27 Intent-to-treat population 28 Intent-to-treat Population 29 Intent-to-treat Population 29 Intent-to-treat Population 29 Intent-to-treat Population 20, 3, 6, 9, 12, 24 Intent-to-treat Population 20, 3, 6, 9, 12, 24 Intent-to-treat Population 26 Intent-to-treat Population 27 Intent-to-treat Population 27 Intent-to-treat Population 29 Intent-to-treat Population 20, 3, 6, 9, 12, 24 Intent-to-treat Population 20, 3, 6, 9, 12, 24 Intent-to-treat Population 20, 3, 6, 9, 12, 24 Intent-to-treat Population 25 Intent-to-treat Population 26 Intent-to-treat Population 27 Intent-to-treat Population 27 Intent-to-treat Population 29 Intent-to-treat Population 20, 3, 6, 9, 12, 24 Intent-to- | | | | | 24months | | | (median, min, |
| RAID fatigue score 0, 3, 6, 9, 12, 24 Intent-to-treat population 25 Intent-to-treat population 26 Intent-to-treat population 27 Intent-to-treat population 28 Intent-to-treat population 29 Intent-to-treat population 20 Intent-to-treat population 20 Intent-to-treat population 20 Intent-to-treat population 21 Intent-to-treat population 22 Intent-to-treat population 23 Intent-to-treat population 24 Intent-to-treat population 25 Intent-to-treat population 26 Intent-to-treat population 27 Intent-to-treat population 28 Intent-to-treat population 29 Intent-to-treat population 20 Intent-to-treat population 20 Intent-to-treat population 20 Intent-to-treat population 25 Intent-to-treat population 26 Intent-to-treat population 27 Intent-to-treat population 28 Intent-to-treat population 19 Intent-to-treat population 19 Intent-to-treat population 29 Intent-to-treat population 10 Intent-to-treat population 10 Intent-to-treat population 11 Intent-to-treat population 12 Intent-to-treat population 13 Intent-to-treat population 14 Intent-to-treat population 15 Intent-to-treat populat | | | | | | | | max if data are |
| RAID fatigue score 0, 3, 6, 9, 12, Treatment group Continuous 15, 18, 21, 24months 24 Intent-to-treat population Population RAPID3 index score 15, 18, 21, 24 population population Population Popula | | | | | | | | non-normal |
| RAID fatigue score 0, 3, 6, 9, 12, 15, 18, 21, 24 Intent-to-treat population 25 Intent-to-treat population 26 Intent-to-treat population 26 Intent-to-treat population 27 Intent-to-treat population 28 Intent-to-treat population 29 Intent-to-treat population 29 Intent-to-treat population 20 Intent-to-treat | | | | | | | | distributed), n |
| 24 Intent-to-treat (m)HAQ score 0, 3, 6, 9, 12, population 25 Intent-to-treat population 26 Intent-to-treat population 26 Intent-to-treat population 26 Intent-to-treat population 27 Intent-to-treat population 28 Intent-to-treat population 29 Intent-to-treat population 29 Intent-to-treat population 20 Intent-to-treat population 20 Intent-to-treat population 20 Intent-to-treat population 21 Intent-to-treat population 24 Intent group 25 Intent-to-treat population 26 Intent-to-treat population 27 Intent-to-treat population 27 Intent-to-treat population 27 Intent-to-treat population 28 Intent-to-treat population 29 Intent-to-treat population 29 Intent-to-treat population 29 Intent-to-treat population 20 Intent-to-treat po | | | | RAID fatigue score | 0, 3, 6, 9, 12, | Treatment group | | Mean (SD) + |
| 24 Intent-to-treat (m)HAQ score 0, 3, 6, 9, 12, population 25 Intent-to-treat population 26 Intent-to-treat EQ-5D score population 26 Intent-to-treat EQ-5D score population 26 Intent-to-treat population 27 Intent population 26 Intent-to-treat population 26 Intent-to-treat EQ-5D score 27 Intent population 27 Intent population 28 Intent-to-treat population 29 Intent-to-treat population 29 Intent-to-treat population 29 Intent-to-treat population 20 Intent | | | | | 15, 18, 21, | | | 95% CI |
| 24 Intent-to-treat (m)HAQ score 0, 3, 6, 9, 12, population population population (m)HAQ score 15, 18, 21, 24 months 25 Intent-to-treat RAPID3 index score population population (population population population population population (population population population population (population population population population population population (population population population population population population population (population population | | | | | 24months | | | (median, min, |
| 24 Intent-to-treat (m)HAQ score 0, 3, 6, 9, 12, 15, 18, 21, 24 population 15, 18, 21, 24 months 25 Intent-to-treat population 26 Intent-to-treat population 26 Intent-to-treat population 27 population 28 population 29 population 26 Intent-to-treat population 26 Intent-to-treat population 27 population 27 population 27 population 28 population 29 population 29 population 29 population 29 population 20 popu | | | | | | | | max if data are |
| 24 Intent-to-treat (m)HAQ score 0, 3, 6, 9, 12, Treatment group Continuous months 25 Intent-to-treat population Population 0, 3, 6, 9, 12, Population Pop | | | | | | | | non-normal |
| 24 Intent-to-treat population pop | | | | | | | | distributed), n |
| 25 Intent-to-treat RAPID3 index score population 25 Intent-to-treat EQ-5D score population 26 Intent-to-treat population 27 Intent-to-treat population 28 Intent-to-treat EQ-5D score 29 Intent-to-treat population 24 Intent-to-treat EQ-5D score 25 Intent-to-treat EQ-5D score 25 In | (m)HAQ | 24 | Intent-to-treat | (m)HAQ score | 0, 3, 6, 9, 12, | Treatment group | Continuous | Mean (SD) + |
| 25 Intent-to-treat RAPID3 index score 0, 3, 6, 9, 12, population 26 Intent-to-treat population 26 Intent-to-treat population 27 Intent EQ-5D score 28 Intent-to-treat population 28 Intent-to-treat population 29 Intent-to-treat 20 Intent-to-treat population 20 Intent-to-treat 20 Intent-to-treat 21 Intent-to-treat 22 Intent-to-treat 24 Intent-to-treat 24 Intent-to-treat 24 Intent-to-treat 25 Intent-to-treat 25 Intent-to-treat 26 Intent-to-treat 26 Intent-to-treat 26 Intent-to-treat 27 Intent-to-treat 25 I | | | population | | 15, 18, 21, 24 | | | 95% CI |
| 25 Intent-to-treat RAPID3 index score 0, 3, 6, 9, 12, population 15, 18, 21, 24 months 26 Intent-to-treat population EQ-5D score 15, 18, 21, 24 population 15, 18, 21, 24 population 24months | | | | | months | | | (median, min, |
| 25 Intent-to-treat RAPID3 index score 0, 3, 6, 9, 12, population 15, 18, 21, 24 months 26 Intent-to-treat population EQ-5D score 0, 3, 6, 9, 12, population 24months 15, 18, 21, 24months | | | | | | | | max if data are |
| 25 Intent-to-treat RAPID3 index score 0, 3, 6, 9, 12, population 15, 18, 21, 24 months 26 Intent-to-treat EQ-5D score population 24months 15, 18, 21, 24 months 24months 24months | | | | | | | | non-normal |
| 25 Intent-to-treat population RAPID3 index score 15, 18, 21, 24 months 26 Intent-to-treat population EQ-5D score population EQ-5D score 15, 18, 21, 24 months Treatment group O, 3, 6, 9, 12, Treatment group Continuous 15, 18, 21, 24months | | | | | | | | distributed), n |
| population 15, 18, 21, 24 months 26 Intent-to-treat population EQ-5D score 15, 18, 21, 24months 15, 18, 21, 24months | RAPID3 | 25 | Intent-to-treat | RAPID3 index score | 0, 3, 6, 9, 12, | Treatment group | | Mean (SD) + |
| 26 Intent-to-treat EQ-5D score 0, 3, 6, 9, 12, Treatment group Continuous 15, 18, 21, 24months | | | population | | 15, 18, 21, 24 | | | 95% CI |
| 26 Intent-to-treat EQ-5D score 0, 3, 6, 9, 12, Treatment group Continuous 15, 18, 21, 24months | | | | | months | | | (median, min, |
| 26 Intent-to-treat EQ-5D score 0, 3, 6, 9, 12, Treatment group Continuous 15, 18, 21, 24months | | | | | | | | max if data are |
| 26 Intent-to-treat EQ-5D score 0, 3, 6, 9, 12, Treatment group Continuous 15, 18, 21, 24months | | | | | | | | non-normal |
| 26 Intent-to-treat EQ-5D score 0, 3, 6, 9, 12, Treatment group Continuous 15, 18, 21, 24months | | | | | | | | distributed), n |
| 15, 18, 21,<br>24months | EuroQoL | 26 | Intent-to-treat | EQ-5D score | 0, 3, 6, 9, 12, | Treatment group | | Mean (SD) + |
| | | | population | | 15, 18, 21, | | | 95% CI |
| max if data are non-normal distributed), n | | | | | 24months | | | (median, min, |
| non-normal distributed), n | | | | | | | | max if data are |
| distributed), n | | | | | | | | non-normal |
| | | | | | | | | distributed), n |

| Table title | Number | Population | Endpoint | Time points or | Covariates or | Type of variable | Summary |
|---|---|---|---|---|---|---|---|
| | | | | how to conglomerate | subgroups | | statistics |
| 57-symptom list | 27 | Intent-to-treat | Number of symptoms | 0 months | Treatment group | Continuous | Mean (SD) |
| | | population | | | | | (median, min, |
| | | | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |
| | | | Change in number of | 0-24 months | Treatment group | Continuous | (SD) Mean |
| | | | symptoms | | | | (median, min, |
| | | | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |
| Laboratory | 28A+28B | 28A. Intent-to- | Hemoglobin SI unit | 0, 3, 6, 12, 18, | Treatment group | Continuous | Mean change |
| results | | treat | (unit: mmol/L) | 24 months | | | from baseline |
| | | population | | | | | (SD) |
| | | 28B. Safety | | | | | (median, min, |
| | | population | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |
| | | | Hemoglobin original | 0, 3, 6, 12, 18, | Treatment group | Continuous | Mean change |
| | | | unit (unit: mmol/L) | 24 months | | | from baseline |
| | | | | | | | (SD) |
| | | | | | | | (median, min, |
| | | | | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed), n |

| distributed), n | | | | | | | |
|---|---|---|---|---|---|---|---|
| normal | | | | | | | |
| data are non- | | | | | | | |
| min, max if | | | | | | | |
| (SD) (median, | | | | (unit: x10^9/L) | | | |
| from baseline | | | 24 months | unit | | | |
| Mean change | Continuous | Treatment group | 0, 3, 6, 12, 18, | White blood cells SI | | | |
| distributed), n | | | | | | | |
| normal | | | | | | | |
| data are non- | | | | | | | |
| min, max if | | | | | | | |
| (SD) (median, | | | | (unit: fl) | | | |
| from baseline | | | 24 months | unit | | | |
| Mean change | Continuous | Treatment group | 0, 3, 6, 12, 18, | Mean cell volume SI | | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | | | | |
| (median, min, | | | | | | | |
| (SD) | | | | | | | |
| from baseline | | | 24 months | unit (unit: g/dl) | | | |
| Mean change | Continuous | Treatment group | 0, 3, 6, 12, 18, | Hemoglobin original | | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | | | | |
| (median, min, | | | | | | | |
| (SD) | | | | | | | |
| from baseline | | | 24 months | unit (unit: g/L) | | | |
| Mean change | Continuous | Treatment group | 0, 3, 6, 12, 18, | Hemoglobin original | | | |
| SIdlistics | | subgroups | conglomerate | | | | |
| *************************************** | | 5 | <b>b</b> | • | | | |
| Value | Type of variable | Covariates or | Time points or | Endpoint | Population | Number | Table title |

| | | | | Table title |
|---|---|---|---|---|
| | | | | tle |
| | | | | Number |
| | | | | Population |
| White blood cells original unit (unit: c/nl) | White blood cells original unit (unit: /ul) | White blood cells original unit (unit: /nl) | White blood cells original unit (unit: x10^9/L) | Endpoint |
| 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | Time points or how to conglomerate |
| Treatment group | Treatment group | Treatment group | Treatment group | Covariates or subgroups |
| Continuous | Continuous | Continuous | Continuous | Type of variable |
| Mean change from baseline (SD) (median, min, max if data are nonnormal | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Summary<br>statistics |

| distributed). n | | | | | | | |
|---|---|---|---|---|---|---|---|
| data are non- | | | | | | | |
| min, max if | | | | x10^3mm/mm^3) | | | |
| (SD) (median, | | | | (unit: | | | |
| from baseline | | | 24 months | original unit | | | |
| Mean change | Continuous | Treatment group | 0, 3, 6, 12, 18, | White blood cells | | | |
| distributed), n | | | | | | | |
| normal | | | | | | | |
| data are non- | | | | | | | |
| min, max if | | | | | | | |
| (SD) (median, | | | | (unit: n/nl) | | | |
| from baseline | | | 24 months | original unit | | | |
| Mean change | Continuous | Treatment group | 0, 3, 6, 12, 18, | White blood cells | | | |
| distributed), n | | | | | | | |
| normal | | | | | | | |
| data are non- | | | | | | | |
| min, max if | | | | | | | |
| (SD) (median, | | | | (unit: Gpt/L) | | | |
| from baseline | | | 24 months | original unit | | | |
| Mean change | Continuous | Treatment group | 0, 3, 6, 12, 18, | White blood cells | | | |
| distributed), n | | | | | | | |
| normal | | | | | | | |
| data are non- | | | | | | | |
| min, max if | | | | | | | |
| (SD) (median, | | | | (unit: G/L) | | | |
| from baseline | | | 24 months | original unit | | | |
| Mean change | Continuous | Treatment group | 0, 3, 6, 12, 18, | White blood cells | | | |
| Statistics | | subgroups | conglomerate | | | | |
| | . ) | | | | | | |
| Summary | Type of variable | Covariates or | Time points or | Endpoint | Population | Number | Table title |

| distributed), n | | | | | | | |
|---|---|---|---|---|---|---|---|
| normal | | | | | | | |
| data are non- | | | | | | | |
| min, max if | | | | | | | |
| (SD) (median, | | | | x10^3mm/mm^3) | | | |
| from baseline | | | 24 months | unit (unit: | | | |
| Mean change | Continuous | Treatment group | 0, 3, 6, 12, 18, | Neutrophils original | | | |
| distributed), n | | | | | | | |
| normal | | | | | | | |
| data are non- | | | | | | | |
| min, max if | | | | | | | |
| (SD) (median, | | | | | | | |
| from baseline | | | 24 months | unit (unit: x10^9/L) | | | |
| Mean change | Continuous | Treatment group | 0, 3, 6, 12, 18, | Neutrophils original | | | |
| distributed), n | | | | | | | |
| normal | | | | | | | |
| data are non- | | | | | | | |
| min, max if | | | | | | | |
| (SD) (median, | | | | | | | |
| from baseline | | | 24 months | (unit: %) | | | |
| Mean change | Continuous | Treatment group | 0, 3, 6, 12, 18, | Neutrophils relatively | | | |
| distributed), n | | | | | | | |
| normal | | | | | | | |
| data are non- | | | | | | | |
| min, max if | | | | | | | |
| (SD) (median, | | | | | | | |
| from baseline | | | 24 months | (unit: x10^9/L) | | | |
| Mean change | Continuous | Treatment group | 0, 3, 6, 12, 18, | Neutrophils SI unit | | | |
| Statistics | | sangroups | conglomerate | | | | |
| c+++ic+icc | • | | <b>bow +</b> . | • | • | | |
| Summary | Type of variable | Covariates or | Time points or | Endpoint | Population | Number | Table title |

| | | | | | | | | | | | | | | | | | | | | | | | Tab |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | | | | | | | | | | | | | Table title |
| | | | | | | | | | | | | | | | | | | | | | | | Number |
| | | | | | | | | | | | | | | | | | | | | | | • | Population |
| מוווג (מוווג. /מב) | Neutrophils original | | | | unit (unit: c/nl) | Neutrophils original | | | | | | unit (unit: G/L) | Neutrophils original | | | | | | unit (unit: /nl) | Neutrophils original | | - | Endpoint |
| 24 MOIUIS | 0, 3, 6, 12, 18, | | | | 24 months | 0, 3, 6, 12, 18, | | | | | | 24 months | 0, 3, 6, 12, 18, | | | | | | 24 months | 0, 3, 6, 12, 18, | conglomerate | how to | Time points or |
| | Treatment group | | | | | Treatment group | | | | | | | Treatment group | | | | | | | Treatment group | 2000 | subgroups | Covariates or |
| | Continuous | | | | | Continuous | | | | | | | Continuous | | | | | | | Continuous | | | Type of variable |
| (SD) (median, min, max if data are non-normal distributed), n | Mean change | normal<br>distributed), n | data are non- | (SD) (median, | from baseline | Mean change | distributed), n | normal | data are non- | min, max if | (SD) (median, | from baseline | Mean change | distributed), n | normal | data are non- | min, max if | (SD) (median, | from baseline | Mean change | | statistics | Summary |

| | | | | Table title |
|---|---|---|---|---|
| | | | | itle |
| | | | | Number |
| | | | | Population |
| Basophils original unit (unit: /nl) | Basophils original unit (unit: x10^9/L) | Basophils relatively (unit: %) | Basophils SI unit (unit:<br>x10^9/L) | Endpoint |
| 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | Time points or how to conglomerate |
| Treatment group | Treatment group | Treatment group | Treatment group | Covariates or subgroups |
| Continuous | Continuous | Continuous | Continuous | Type of variable |
| Mean change from baseline (SD) (median, min, max if data are nonnormal | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Summary<br>statistics |

| | | | | Table title |
|---|---|---|---|---|
| | | | | Number |
| | | | | Population |
| Eosinophils SI unit<br>(unit: x10^9/L) | Basophils original unit (unit: x10^3mm/mm^3) | Basophils original unit (unit: G/L) | Basophils original unit (unit: /uL) | Endpoint |
| 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | Time points or how to conglomerate |
| Treatment group | Treatment group | Treatment group | Treatment group | Covariates or subgroups |
| Continuous | Continuous | Continuous | Continuous | Type of variable |
| Mean change from baseline (SD) (median, min, max if data are nonnormal | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Summary<br>statistics |

| | | | | Table title |
|---|---|---|---|---|
| | | | | title |
| | | | | Number |
| | | | | Population |
| Eosinophils original<br>unit (unit: G/L) | Eosinophils original unit (unit: /uL) | Eosinophils original unit (unit: /nl) | Eosinophils relatively (unit: %) | Endpoint |
| 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | Time points or how to conglomerate |
| Treatment group | Treatment group | Treatment group | Treatment group | Covariates or subgroups |
| Continuous | Continuous | Continuous | Continuous | Type of variable |
| Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Summary<br>statistics |

| | | | | Table title |
|---|---|---|---|---|
| | | | | ति |
| | | | | Number |
| | | | | Population |
| Lymphocytes original unit (unit: x10^9/L) | Lymphocytes relatively (unit: %) | Lymphocytes SI unit<br>(unit: x10^9/L) | Eosinophils original unit (unit: x10^3mm/mm^3) | Endpoint |
| 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | Time points or how to conglomerate |
| Treatment group | Treatment group | Treatment group | Treatment group | Covariates or subgroups |
| Continuous | Continuous | Continuous | Continuous | Type of variable |
| Mean change from baseline (SD) (median, min, max if data are nonnormal | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Summary<br>statistics |

| distributed), n | | | | | | | |
|---|---|---|---|---|---|---|---|
| normal | | | | | | | |
| data are non- | | | | | | | |
| min, max if | | | | | | | |
| (SD) (median, | | | | | | | |
| from baseline | | | 24 months | unit (unit: G/L) | | | |
| Mean change | Continuous | Treatment group | 0, 3, 6, 12, 18, | Lymphocytes original | | | |
| distributed), n | | | | | | | |
| normal | | | | | | | |
| data are non- | | | | | | | |
| min, max if | | | | | | | |
| (SD) (median, | | | | | | | |
| from baseline | | | 24 months | unit (unit: c/nl) | | | |
| Mean change | Continuous | Treatment group | 0, 3, 6, 12, 18, | Lymphocytes original | | | |
| distributed), n | | | | | | | |
| normal | | | | | | | |
| data are non- | | | | | | | |
| min, max if | | | | | | | |
| (SD) (median, | | | | | | | |
| from baseline | | | 24 months | unit (unit: /uL) | | | |
| Mean change | Continuous | Treatment group | 0, 3, 6, 12, 18, | Lymphocytes original | | | |
| distributed), n | | | | | | | |
| normal | | | | | | | |
| data are non- | | | | | | | |
| min, max if | | | | | | | |
| (SD) (median, | | | | | | | |
| from baseline | | | 24 months | unit (unit: /nl) | | | |
| Mean change | Continuous | Treatment group | 0, 3, 6, 12, 18, | Lymphocytes original | | | |
| Statistics | | sabgroups | conglomerate | | | | |
| 1 | | | <b>b</b> | - | - | | |
| Summary | Type of variable | Covariates or | Time points or | Endpoint | Population | Number | Table title |

| distributed) n | | | | | | | |
|---|---|---|---|---|---|---|---|
| normal | | | | | | | |
| data are non- | | | | | | | |
| min, max if | | | | | | | |
| (SD) (median, | | | | | | | |
| from baseline | | | 24 months | unit (unit: x10^9/L) | | | |
| Mean change | Continuous | Treatment group | 0, 3, 6, 12, 18, | Monocytes original | | | |
| distributed), n | | | | | | | |
| normal | | | | | | | |
| data are non- | | | | | | | |
| min, max if | | | | | | | |
| (SD) (median, | | | | | | | |
| from baseline | | | 24 months | (unit: %) | | | |
| Mean change | Continuous | Treatment group | 0, 3, 6, 12, 18, | Monocytes relatively | | | |
| distributed), n | | | | | | | |
| normal | | | | | | | |
| data are non- | | | | | | | |
| min, max if | | | | | | | |
| (SD) (median, | | | | | | | |
| from baseline | | | 24 months | (unit: x10^9/L) | | | |
| Mean change | Continuous | Treatment group | 0, 3, 6, 12, 18, | Monocytes SI unit | | | |
| distributed), n | | | | | | | |
| normal | | | | | | | |
| data are non- | | | | | | | |
| min, max if | | | | | | | |
| (SD) (median, | | | | x10^3mm/mm^3) | | | |
| from baseline | | | 24 months | (unit: | | | |
| Mean change | Continuous | Treatment group | 0, 3, 6, 12, 18, | Lymphocytes | | | |
| | | 0.00 | conglomerate | | | | |
| statistics | | subgroups | how to | | , | | |
| Summary | Type of variable | Covariates or | Time points or | Endpoint | Population | Number | Table title |

| | | | | Table title |
|---|---|---|---|---|
| | | | | itle |
| | | | | Number |
| | | | | Population |
| Monocytes original unit (unit: x10^3mm/mm^3) | Monocytes original unit (unit: G/L) | Monocytes original unit (unit: /uL) | Monocytes original unit (unit: /nl) | Endpoint |
| 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | Time points or how to conglomerate |
| Treatment group | Treatment group | Treatment group | Treatment group | Covariates or subgroups |
| Continuous | Continuous | Continuous | Continuous | Type of variable |
| Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Summary<br>statistics |

| | | | | Table title |
|---|---|---|---|---|
| | | | | title |
| | | | | Number |
| | | | | Population |
| Platelets original unit (unit: /uL) | Platelets original unit (unit: /nl) | Platelets original unit<br>(unit: x10^9/L) | Platelets SI unit<br>(unit: x10^9/L) | Endpoint |
| 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | Time points or how to conglomerate |
| Treatment group | Treatment group | Treatment group | Treatment group | Covariates or subgroups |
| Continuous | Continuous | Continuous | Continuous | Type of variable |
| Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Summary<br>statistics |

| | | | | Table |
|---|---|---|---|---|
| | | | | Table title |
| | | | | Number |
| | | | | Population |
| Platelets original unit<br>(unit: 10^3mm/mm^3) | Platelets original unit<br>(unit: Gpt/L) | Platelets original unit<br>(unit: G/L) | Platelets original unit (unit: c/nl) | Endpoint |
| 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | Time points or how to conglomerate |
| Treatment group | Treatment group | Treatment group | Treatment group | Covariates or subgroups |
| Continuous | Continuous | Continuous | Continuous | Type of variable |
| Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Summary<br>statistics |

| | | | | Table title |
|---|---|---|---|---|
| | | | | Number |
| | | | | Population |
| Creatinine SI unit<br>(unit: mcmol/L) | Glucose original unit<br>(unit: mg/dl) | Glucose original unit<br>(unit: mmol/L) | Glucose SI unit<br>(unit: mmol/L) | Endpoint |
| 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | Time points or how to conglomerate |
| Treatment group | Treatment group | Treatment group | Treatment group | Covariates or subgroups |
| Continuous | Continuous | Continuous | Continuous | Type of variable |
| Mean change from baseline (SD) (median, min, max if data are nonnormal distributed). n | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Summary<br>statistics |

| 1011-110111101 | | | | | | | |
|---|---|---|---|---|---|---|---|
| non-normal | | | | | | | |
| max if data are | | | | | | | |
| (median, min, | | | | | | | |
| (SD) | | | | | | | |
| from baseline | | | 24 months | (unit: mg/dl) | | | |
| Mean change | Continuous | Treatment group | 0, 3, 6, 12, 18, | Creatinine original unit | | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | | | | |
| (median, min, | | | | | | | |
| (SD) | | | | | | | |
| from baseline | | | 24 months | (unit: mcmol/L) | | | |
| Mean change | Continuous | Treatment group | 0, 3, 6, 12, 18, | Creatinine original unit | | | |
| | | | conglomerate | | | | |
| statistics | | subgroups | how to | | | | |
| Summary | Type of variable | Covariates or | Time points or | Endpoint | Population | Number | Table title |
| , | _ , | | • | | T | -<br>: | |

| | | | | Table title |
|---|---|---|---|---|
| | | | | itle |
| | | | | Number |
| | | | | Population |
| Cholesterol SI unit<br>(unit: mmol/L) | ALAT original unit (unit: umol/s*I) | ALAT original unit<br>(unit: ukat/L) | ALAT original unit<br>(unit: U/L) | Endpoint |
| 0, 3, 12, 24<br>months | 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | 0, 3, 6, 12, 18,<br>24 months | Time points or how to conglomerate |
| Treatment group | Treatment group | Treatment group | Treatment group | Covariates or subgroups |
| Continuous | Continuous | Continuous | Continuous | Type of variable |
| Mean change from baseline (SD) (median, min, max if data are nonnormal | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Summary<br>statistics |

| distributed), n | | | | | | | |
|---|---|---|---|---|---|---|---|
| normal | | | | | | | |
| data are non- | | | | | | | |
| min, max if | | | | | | | |
| (SD) (median, | | | | (unit: mmol/L) | | | |
| from baseline | | | months | original unit | | | |
| Mean change | Continuous | Treatment group | 0, 3, 12, 24 | HDL cholesterol | | | |
| distributed), n | | | | | | | |
| normal | | | | | | | |
| data are non- | | | | | | | |
| min, max if | | | | | | | |
| (SD) (median, | | | | | | | |
| from baseline | | | months | (unit: mmol/L) | | | |
| Mean change | Continuous | Treatment group | 0, 3, 12, 24 | HDL cholesterol SI unit | 1 | | |
| distributed), n | | | | | | | |
| normal | | | | | | | |
| data are non- | | | | | | | |
| min, max if | | | | | | | |
| (SD) (median, | | | | | | | |
| from baseline | | | months | unit (unit: mg/dl) | | | |
| Mean change | Continuous | Treatment group | 0, 3, 12, 24 | Cholesterol original | | | |
| distributed), n | | | | | | | |
| normal | | | | | | | |
| data are non- | | | | | | | |
| min, max if | | | | | | | |
| (SD) (median, | | | | | | | |
| from baseline | | | months | unit (unit: mmol/L) | | | |
| Mean change | Continuous | Treatment group | 0, 3, 12, 24 | Cholesterol original | | | |
| SIGUSTICS | | sabgroups | conglomerate | | | | |
| ********* | | | <b>b</b> | | | | |
| Value | Type of variable | Covariates or | Time points or | Endpoint | Population | Number | Table title |
| | | | | | | 1 | |

| | | | | Table title |
|---|---|---|---|---|
| 29A + 29B | | | | Number |
| 29A. Intent-to-<br>treat<br>population<br>29B. Safety<br>population | | | | Population |
| Weight (kg) | ESR SI unit<br>(unit: mm/h) | CRP SI unit<br>(unit: mg/L) | HDL cholesterol<br>original unit<br>(unit: mg/dl) | Endpoint |
| 0, 3, 6, 12, 18,<br>24months | 0, 3, 6, 12, 18,<br>24, 27 months | 0, 3, 6, 12, 18,<br>24, 27 months | 0, 3, 12, 24<br>months | Time points or how to conglomerate |
| Treatment group | Treatment group | Treatment group | Treatment group | Covariates or subgroups |
| Continuous | Continuous | Continuous | Continuous | Type of variable |
| Mean change from baseline (SD) (median, min, max if data are non-normal | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Mean change from baseline (SD) (median, min, max if data are nonnormal distributed), n | Summary<br>statistics |

| distributed), n | | | | | | | |
|---|---|---|---|---|---|---|---|
| normal | | | | | | | |
| data are non- | | | | | | | |
| min, max if | | | | | | | |
| (SD) (median, | | | | | | | |
| from baseline | | | 24 months | | | | |
| Mean change | Continuous | Treatment group | 0, 3, 6, 12, 18, | Heart rate per minute | | | |
| distributed), n | | | | | | | |
| normal | | | | | | | |
| data are non- | | | | | | | |
| min, max if | | | | | | | |
| (SD) (median, | | | | | | | |
| from baseline | | | 24 months | pressure (mmHg) | | | |
| Mean change | Continuous | Treatment group | 0, 3, 6, 12, 18, | Diastolic blood | | | |
| distributed), n | | | | | | | |
| normal | | | | | | | |
| data are non- | | | | | | | |
| min, max if | | | | | | | |
| (SD) (median, | | | | | | | |
| from baseline | | | 24 months | pressure (mmHg) | | | |
| Mean change | Continuous | Treatment group | 0, 3, 6, 12, 18, | Systolic blood | | | |
| distributed), n | | | | | | | |
| normal | | | | | | | |
| data are non- | | | | | | | |
| min, max if | | | | | | | |
| (SD) (median, | | | | | | | |
| from baseline | | | | | | | |
| Mean change | Continuous | Treatment group | 0, 24 months | Height (cm) | | | |
| | | 0.00 | conglomerate | | | | |
| statistics | | subgroups | how to | | | | |
| Summary | Type of variable | Covariates or | Time points or | Endpoint | Population | Number | Table title |

| non-normal | | | | | | | |
|---|---|---|---|---|---|---|---|
| max if data are | | | | caps | | | |
| (median, min, | | | months | according to electronic | population | | |
| Mean (SD) | Continuous | Treatment group | 3, 6, 12, 18, 24 | % adherence | Safety | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | | | | |
| (median, min, | | | months | according to pill count | population | | |
| Mean (SD) | Continuous | Treatment group | 3, 6, 12, 18, 24 | % adherence | Safety | 30C | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | caps | | | |
| (median, min, | | | | according to electronic | population | | |
| Mean (SD) | Continuous | Treatment group | 3 months | % adherence | Per-protocol | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | | | | |
| (median, min, | | | | according to pill count | population | | |
| Mean (SD) | Continuous | Treatment group | 3 months | % adherence | Per-protocol | 30B | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | caps | | | |
| (median, min, | | | months | according to electronic | population | | |
| Mean (SD) | Continuous | Treatment group | 3, 6, 12, 18, 24 | % adherence | Intent-to-treat | | |
| distributed), n | | | | | | | |
| non-normal | | | | | | | |
| max if data are | | | | | | | |
| (median, min, | | | months | according to pill count | population | | |
| Mean (SD) | Continuous | Treatment group | 3, 6, 12, 18, 24 | % adherence | Intent-to-treat | 30A | Adherence |
| | | 0 7 | conglomerate | | | | |
| statistics | : | subgroups | how to | | • | | |
| Summary | Type of variable | Covariates or | Time points or | Endpoint | Population | Number | Table title |

| <b>ナ</b> _ | N1 | 7 - ;; l _ L ! | 7 | 1: | ) | | · |
|---|---|---|---|---|---|---|---|
| ומטופ נונופ | Nulliber | Population | Enapoint | illie politis of | COVALIATES OF | Type of variable | Summary |
| | | | | conglomerate | subgroups | | SIdlibiles |
| Concomitant | 31 | Intent-to-treat | Concomitant | Baseline | Treatment group | Dichotomous/continuous | -DMARDs: % |
| medications | | population | medication summary | | | | (n) |
| summary | | | | | | | -NSAIDs: % (n) |
| | | | | | | | -Biologicals: % |
| | | | | | | | (n) |
| | | | | | | | -Other anti- |
| | | | | | | | rheumatic |
| | | | | | | | medication: % |
| | | | | | | | (n) |
| | | | | | | | -Other |
| | | | | | | | medication: |
| | | | | | | | Mean number |
| | | | | | | | (SD) (median, |
| | | | | | | | min, max if |
| | | | | | | | data are non- |
| | | | | | | | normal |
| | | | | | | | distributed) |
| | | | | | | | -Top 3 of most |
| | | | | | | | common |
| | | | | | | | concomitant |
| | | | | | | | medication |
| | | | | | | | class: |
| | | | | | | | 1. % (n) |
| | | | | | | | 2. % (n) |
| | | | | | | | 3. % (n) |

| Intent-to-treat Bone mass lumber 0, 24 months Treatment group Continuous population population Intent-to-treat Change in bone mass hip population intent-to-treat Change in bone mass hip population intent-to-treat Change in bone mass population intent-to-treat Change in bone mass population hip population with at least one incident compression fracture (by VFA or lateral spine films). | Table title | Number | Population | Endpoint | Time points or | Covariates or | Type of variable | Summary |
|---|---|---|---|---|---|---|---|---|
| 32 Intent-to-treat population Spine Sp | | | | | how to conglomerate | subgroups | | statistics |
| eat Change in bone mass O-24 months Treatment group Continuous eat Change in bone mass hip O, 24 months Treatment group Continuous eat Change in bone mass O-24 months Treatment group Continuous hip Treatment group Continuous Treatment group Continuous Treatment group Continuous Treatment group Continuous Treatment group Dichotomous incident compression fracture (by VFA or lateral spine films) | Bone mass | 32 | Intent-to-treat | Bone mass lumber | 0, 24 months | Treatment group | | Mean (SD) + |
| reat Change in bone mass 0-24 months Treatment group Continuous reat Bone mass hip 0, 24 months Treatment group Continuous reat Change in bone mass 0-24 months Treatment group Continuous hip Continuous Treatment group Continuous Treatment group Dichotomous with at least one incident compression fracture (by VFA or lateral spine films) Treatment group Dichotomous | | | population | spine | | | | 95% CI |
| reat Change in bone mass | | | | | | | | max if data are |
| reat Change in bone mass 0-24 months Treatment group Continuous reat Bone mass hip 0, 24 months Treatment group Continuous reat Change in bone mass 0-24 months Treatment group Continuous hip Continuous Treatment group Continuous Treatment group Continuous Treatment group Continuous Treatment group Continuous Treatment group Dichotomous with at least one incident compression fracture (by VFA or lateral spine films) | | | | | | | | non-normal |
| reat Change in bone mass 0-24 months Treatment group Continuous reat Bone mass hip 0, 24 months Treatment group Continuous reat Change in bone mass 0-24 months Treatment group Continuous reat Change in bone mass 0-24 months Treatment group Continuous hip Continuous reat Number of patients 24 months Treatment group Dichotomous with at least one incident compression fracture (by VFA or lateral spine films) lateral spine films) Treatment group Dichotomous Treatme | | | | | | | | distributed), n |
| eat Bone mass hip 0, 24 months Treatment group Continuous eat Change in bone mass 0-24 months Treatment group Continuous hip eat Number of patients with at least one incident compression fracture (by VFA or lateral spine films) Treatment group Dichotomous Dichotomous | | | Intent-to-treat | Change in bone mass | 0-24 months | Treatment group | | Mean (SD) + |
| reat Bone mass hip 0, 24 months Treatment group Continuous reat Change in bone mass 0-24 months Treatment group Continuous reat Number of patients with at least one incident compression fracture (by VFA or lateral spine films) Treatment group Dichotomous Dichotomous | | | population | lumbar spine | | | | 95% CI |
| reat Bone mass hip 0, 24 months Treatment group Continuous reat Change in bone mass 0-24 months Treatment group Continuous hip reat Number of patients with at least one incident compression fracture (by VFA or lateral spine films) Treatment group Dichotomous Dichotomous | | | | | | | | (median, min, |
| reat Bone mass hip 0, 24 months Treatment group Continuous reat Change in bone mass 0-24 months Treatment group Continuous hip reat Number of patients with at least one incident compression fracture (by VFA or lateral spine films) Treatment group Dichotomous Dichotomous | | | | | | | | max if data are |
| reat Bone mass hip 0, 24 months Treatment group Continuous reat Change in bone mass 0-24 months Treatment group Continuous hip reat Number of patients with at least one incident compression fracture (by VFA or lateral spine films) Treatment group Dichotomous Dichotomous | | | | | | | | non-normal |
| reat Change in bone mass D-24 months Treatment group Continuous hip Treatment group Continuous Continuous Preat Change in bone mass Preatment group Continuous Continuous Preatment group With at least one incident compression fracture (by VFA or lateral spine films) Treatment group Dichotomous Preatment group Preatm | | | | | | | | distributed), n |
| reat Change in bone mass 0-24 months Treatment group Continuous hip The atment group Continuous The atment group Continuous Treatment group Dichotomous With at least one incident compression fracture (by VFA or lateral spine films) | | | Intent-to-treat | Bone mass hip | 0, 24 months | Treatment group | Continuous | Mean (SD) + |
| reat Change in bone mass 0-24 months Treatment group Continuous hip Treatment group Continuous Treatment group Dichotomous With at least one incident compression fracture (by VFA or lateral spine films) | | | population | | | | | 95% CI |
| reat Change in bone mass 0-24 months Treatment group Continuous hip Treatment group Continuous | | | | | | | | (median, min, |
| reat Change in bone mass 0-24 months Treatment group Continuous hip Treatment group Continuous Treatment group Dichotomous with at least one incident compression fracture (by VFA or lateral spine films) | | | | | | | | max if data are |
| reat Change in bone mass 0-24 months Treatment group Continuous hip reat Number of patients with at least one incident compression fracture (by VFA or lateral spine films) Treatment group Dichotomous Treatment group Dichotomous | | | | | | | | non-normal |
| reat Change in bone mass 0-24 months Treatment group Continuous hip reat Number of patients with at least one incident compression fracture (by VFA or lateral spine films) Treatment group Dichotomous Treatment group Dichotomous | | | | | | | | distributed), n |
| reat Number of patients 24 months Treatment group Dichotomous incident compression fracture (by VFA or lateral spine films) | | | Intent-to-treat | Change in bone mass | 0-24 months | Treatment group | | Mean (SD) + |
| reat Number of patients 24 months Treatment group Dichotomous with at least one incident compression fracture (by VFA or lateral spine films) | | | population | hip | | | | 95% CI |
| reat Number of patients 24 months Treatment group Dichotomous with at least one incident compression fracture (by VFA or lateral spine films) | | | | | | | | (median, min, |
| reat Number of patients 24 months Treatment group Dichotomous with at least one incident compression fracture (by VFA or lateral spine films) | | | | | | | | max if data are |
| reat Number of patients 24 months Treatment group Dichotomous with at least one incident compression fracture (by VFA or lateral spine films) | | | | | | | | non-normal |
| reat Number of patients 24 months Treatment group Dichotomous with at least one incident compression fracture (by VFA or lateral spine films) | | | | | | | | מוזנווטמנכט), וו |
| | | | Intent-to-treat | Number of patients | 24 months | Treatment group | Dichotomous | % (n), yes |
| incident compression fracture (by VFA or lateral spine films) | | | population | with at least one | | | | |
| fracture (by VFA or lateral spine films) | | | | incident compression | | | | |
| lateral spine films) | | | | fracture (by VFA or | | | | |
| | | | | lateral spine films) | | | | |

| | | | | | | | 0 - 7 |
|---|---|---|---|---|---|---|---|
| | | | 15, 18, 21, 24<br>months | replacement surgeries | population | | replacement |
| | Continuous | Treatment group | 0, 3, 6, 9, 12, | Number of joint | Intent-to-treat | 35 | Joint |
| | | | | fractures | | | fractures |
| | | | | vertebrae with | | | vertebrae with |
| | | | | height loss in | population | | height loss in |
| | Continuous | Treatment group | 0- months | Distribution of % | Intent-to-treat | 34 | Distribution of % |
| | | | | | | | films) |
| | | | | | | | or lateral spine |
| | | | | | | | fractures (by VFA |
| | | | | | | | vertebral |
| | | | | vertebral fractures | population | | prevalent |
| | Continuous | Treatment group | 0 months | Number of prevalent | Intent-to-treat | 33 | Number of |
| | | | | spine films) | | | |
| | | | | (by VFA or lateral | | | |
| | | | | compression fractures | population | | |
| | Continuous | Treatment group | 24 months | Number of incident | Intent-to-treat | | |
| | | | conglomerate | | | | |
| | | subgroups | how to | | | | |
| le | Type of variable | Covariates or | Time points or | Endpoint | Population | Number | Table title |

| 4-1,1, 1;11, | N1 L | 7latia | 7: L: )::+ | 1 | ) | # | |
|---|---|---|---|---|---|---|---|
| ומטוכ נונות | | רסקמומוסוו | רומקסוור | how to | subgroups | י אָבר כו אמו מצות | statistics |
| AE, SAE, other AE | 36A | Intent-to-treat | Number of AEs, SAEs, | 3, 24 months | Treatment group | Continuous | -Mean (SD) |
| of special | | population | other AEs of special | | | | (median, min, |
| summary | | | IIIterest | | | | non-normal |
| , | | | | | | | distributed) |
| | | | | | | | -Top 3 of most |
| | | | | | | | common AE |
| | | | | | | | categories: |
| | | | | | | | 1. % (n) |
| | | | | | | | 2. % (n) |
| | | | | | | | 3. % (n) |
| | 36B | Safety | Number of AEs, SAEs, | 3, 24 months | Treatment group | Continuous | -Mean (SD) |
| | | population | other AEs of special | | | | (median, min, |
| | | | Interest | | | | max if data are |
| | | | | | | | non-normal |
| | | | | | | | distributed) |
| | | | | | | | -Top 3 of most |
| | | | | | | | common AE |
| | | | | | | | categories: |
| | | | | | | | 1. % (n) |
| | | | | | | | 2. % (n) |
| | | | | | | | 3. % (n) |
| AEs, SAEs, other | 36C | Intent-to-treat | Number of AE, SAE, | 3, 24 months | Treatment group | Categorical | -Category 1: n |
| AEs of special | | population | other AE of special | | | | (%) |
| interest | | | interest per organ | | | | -Category 2: |
| | | | system | | | | (n%) |
| | | | | | | | -Category 3: n |
| | | | | | | | (%) |
| | | | | | | | Etc. |
| Table title | Number | Population | Endpoint | Time points or | Covariates or | Type of variable | Summary |
|---|---|---|---|---|---|---|---|
| | | | | how to | subgroups | | statistics |
| | | | | conglomerate | | | |
| | 36D | Safety | Number of AE, SAE, | 3, 24 months | Treatment group | Categorical | -Category 1: n |
| | | population | other AE of special | | | | (%) |
| | | | interest per organ | | | | -Category 2: |
| | | | system | | | | (n%) |
| | | | | | | | -Category 3: n |
| | | | | | | | (%) |
| | | | | | | | Etc. |
| Presence of SAE | 37 | Intent-to-treat | Presence of SAE or | 24 months | Treatment group | Dichotomous | -Yes: n(%) |
| or other AE of | | population | other AE of special | | | | -No: n(%) |
| special interest | | | interest | | | | |

| Figure 1 | Patient disposition: consort flow chart |
|---|---|
| Figure 2 | Premature discontinuation per treatment group: Kaplan-Meier survival curve |
| Figure 2 | DAS28 score per treatment group over time |
| Figure 3 | Number of SAEs and other AEs of special interest per treatment group: Kaplan-Meier survival curve |
| Figure 4 | Probability density plot of x-rays at 0 and 24 months |

| Listing 1 | Patient disposition |
|---|---|
| Listing 2 | Patients excluded from the analysis populations |
| Listing 3 | Protocol violations |
| Listing 4 | Visit windows |
| Listing 5 | Study completion including reason early withdrawal |
| Listing 6 | Demographics and baseline characteristics |
| Listing 7 | History of glaucoma and cataract |
| Listing 8 | RA history |
| Listing 9.A | Medical history |
| Listing 9.B | Medical history with MedDRA Coding |
| Listing 10.A | Treatment not given according to protocol - interrupted |
| Listing 10.B | Treatment not given according to protocol – discontinued |
| Listing 11 | Change of antirheumatic treatment, with reason |
| Listing 12<br>Listing 13 | Intensification of treatment for existing comorbidity, e.g. hypertension or diabetes DAS28 scores, DAS44 scores and EULAR response |
| Listing 14 | Swollen and tender joints |
| Listing 15.A | Patient global assessment of disease |
| Listing 15.B | Physician global assessment of disease |
| Listing 16 | ACR 20 response |
| Listing 17 | Minimal disease activity |
| Listing 18 | Total Sharp/van der Heijde damage score of hands and forefeet radiographs |
| Listing 19 | Morning stiffness |
| Listing 20.A | SF-36 questionnaire |
| Listing 20.B | SF-36 scores |
| Listing 21.A | (m)HAQ questionnaire |
| Listing 21.B | (m)HAQ scores |
| Listing 22.A | RAID questionnaire |
| Listing 22.B | RAID scores |
| Listing 23.A | EQ-5D questionnaire |
| Listing 23.B | EQ-5D scores |
| Listing 24 | Patient symptom list questionnaire |
| Listing 25.A | Laboratory – Hematology and chemistry |
| Listing 25.B | Laboratory – Lipids |
| Listing 25.C | Laboratory – CRP and ESR |
| Listing 26 | Vital signs |
| Listing 27 | Physical examination |
| Listing 28 | Previous medication |
| Listing 29 | Concomitant medications |
| Listing 30.A | Adverse events |
| Listing 30.B | Serious adverse events |
| Listing 30.C | Other adverse events of special interest |
| Listing 31 | Death |

## 8 Statistical software

The statistical programming and analysis platform R will be used for the analysis (R Core Team, 2020).

SPSS version 26 or higher will be used for the descriptive statistics. Graphpad Prism version 9.0.2 or higher will be used for the figures.

# 9 References

Aletaha D, Neogi T, Silman AJ, et al. 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum. 2010 Sep;62(9):2569-81.

Bakker MF, Jacobs JW, Welsing PM, et al. Low-dose prednisone inclusion in a methotrexate-based, tight control strategy for early rheumatoid arthritis: a randomized trial. Annals of Internal Medicine 2012;156:329-39.

Benjamini Y, Hochberg Y. Controlling the False Discovery Rate: A Practical and Powerful Approach to Multiple Testing. Journal of the Royal Statistical Society Series B (Methodological) 1995;57:289-300.

Buttgereit F, Mehta D, Kirwan J, Szechinski J, Boers M, Alten RE, et al. Low-dose prednisone chronotherapy for rheumatoid arthritis: a randomised clinical trial (CAPRA-2). Ann Rheum Dis 2013;72:204-10.

Felson DT, Anderson JJ, Boers M, Bombardier C, Furst D, Goldsmith C, et al. American College of Rheumatology. Preliminary definition of improvement in rheumatoid arthritis. Arthritis Rheum 1995 Jun;38(6):727-35.

Felson DT, Smolen JS, Wells G, Zhang B, van Tuyl LH, Funovits J, et al. American College of Rheumatology/European League against Rheumatism provisional definition of remission in rheumatoid arthritis for clinical trials. Ann Rheum Dis 2011;70:404-13.

Genant HK, Jergas M, Palermo L, Nevitt M, Valentin RS, Black D, et al. Comparison of semiquantitative visual and quantitative morphometric assessment of prevalent and incident vertebral fractures in osteoporosis The Study of Osteoporotic Fractures Research Group. J Bone Miner Res 1996;11:984-96.

Guyatt GH, Norris SL, Schulman S, Hirsh J, Eckman MH, Akl EA, et al. American College of Chest Physicians. Methodology for the development of antithrombotic therapy and prevention of thrombosis guidelines: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):53S-70S.

Hox JJ. Multilevel analysis. Techniques and applications. New York: Routledge; 2010.

Kuznetsova A, Brockhoff PB, Christensen RHB. ImerTest Package: Tests in Linear Mixed Effects Models.J Stat Softw 2017;82:1-26. https://doi.org/10.18637/jss.v082.i13

Little RJA, Rubin DB. Statistical analysis with missing data (2nd ed.). Hoboken: Wiley; 2002.

R Core Team. R: A language and environment for statistical computing. Vienna; R Foundation for Statistical Computing; 2020. https://www.R-project.org/

Ritchie DM, Boyle JA, McInnes JM et al. Clinical studies with an articular index for the assessment of joint tenderness in patients with rheumatoid arthritis. Q J Med 1968; 37: 393-406.

Rubin DB. Causal Inference Using Potential Outcomes. J Am Stat Assoc 2005;100:322-31. http://doi.org/10.1198/016214504000001880

Sharp JT, Young DY, Bluhm GB et al. How many joints in the hands and wrists should be included in a score of radiologic abnormalities used to assess rheumatoid arthritis? Arthritis Rheum 1985; 28: 1326-35.

Snijders TAB, Bosker RJ. Multilevel Analysis: An Introduction to Basic and Advanced Multilevel Modeling. New York: SAGE; 2011.

Van Buuren S. Flexible Imputation of Missing Data. Boca Raton: CRC Press; 2012.

Van der Heijde DM, Van Riel P, Nuver-Zwart IH, Gribnau FW, Van der Putte LB. Effects of hydroxychloroquine and sulphasalazine on progression of joint damage in rheumatoid arthritis. Lancet 1989; 1: 1036-8.

Van Gestel AM, Prevoo ML, Van 't Hof MA, Van Rijswijk MH, Van de Putte LB, Van Riel PL. Development and validation of the European League Against Rheumatism response criteria for rheumatoid arthritis. Comparison with the preliminary American College of Rheumatology and the World Health Organization/International League Against Rheumatism Criteria. Arthritis Rheum. 1996 Jan;39(1):34-40.

Van Gestel AM, Anderson JJ, Van Riel PL, Boers M, Haagsma CJ, Rich B, Wells G, Lange ML, Felson DT. ACR and EULAR improvement criteria have comparable validity in rheumatoid arthritis trials. American College of Rheumatology European League of Associations for Rheumatology. J Rheumatol. 1999 Mar;26(3):705-11.

Wells, G.A., Boers, M., Shea, B., Brooks, P.M., Simon, L.S., Strand, C.V., et al. (2005). Minimal disease activity for rheumatoid arthritis: a preliminary definition. J Rheumatol, 32, 2016-24.

# 10 Appendix A: secondary outcome measures that need further specification

# Remission and minimal disease activity (MDA), according to ACR/EULAR criteria

Remission is defined according to the Boolean Based definition of remission in clinical trials. A patient must satisfy a tender joint count  $\leq 1$ , a swollen joint count  $\leq 1$ , CRP  $\leq 1$  mg/dL, and a patient global assessment  $\leq 1$  (on a 0-10 scale). MDA is defined as a DAS28 < 2.6 (Felson et al., 2011; Wells et al., 2005).

## **ACR** response

This index is described in the protocol. To calculate ACR50 and 70, the '20%' criterion is replaced by 50 resp 70%.

## Vital signs

Systolic and diastolic blood pressure, pulse rate, weight and height.

# **Physical examinations**

Physical examinations were performed at the discretion of the treating physician. The results will be summarized in a table per treatment group. All abnormalities will be reported.

#### Bone mass assessment

Bone mass of lumbar spine and total hip is assessed by Dual-energy X-ray Absorptiometry (DEXA), and expressed as g/cm<sup>2</sup> for analysis.

In addition, description of bone mass at femoral neck, and bone mass of all sites as T-score.

# Vertebral fracture analysis (by DEXA, or alternatively, by assessment of lateral spine X-rays)

Vertebrae are viewed on transversal image and height loss (%) is scored according to Genant:

Grade 0: <20%; Grade 1: 20-25%; Grade 2 ≥25-40%; Grade 3 >40%.

baseline: prevalent fracture: number of vertebrae with at least Grade 1;

description of distribution of % height loss in vertebrae of patients with a prevalent fracture.

follow up: incident fracture: sum of:

a. number of vertebrae with baseline Grade 0 increasing to Grade 1-3

(% height loss <20% increasing to >20%)

b. number of vertebrae with baseline Grade >0 increasing in Grade

(Grade 1 increasing to 2 or 3; Grade 2 increasing to 3)

## **Medication adherence**

Medication adherence according to pill count is calculated as follows: if the number of capsules dispensed is D, the treatment period in number of days is P, and the number of capsules returned is R, medication adherence (expressed as %) is calculated as: 100\*(D-R)/P. In alignment with the literature, good medication adherence is defined as an intake of at least 80% of the prescribed doses.

For medication adherence according to electronic caps the assumption is made that a bottle opening is equal to the intake of one capsule. If the number of days that the cap wis not opened is O and the treatment period in number of days is P, adherence according to electronic caps (expressed as %) is calculated as: 100\*(P-O)/P.

# 11 Appendix B – Modifications from the protocol

#### **Definition of AESI**

We refined the definitions of AESI in the protocol because it was not always completely clear when we were adjudicating the blinded events. The protocol text has been updated in order to make binding decisions on whether an event is AESI or not. The following changes and clarifications to the definition of an AESI were made:

- 'Stop of antirheumatic treatment for AE' was one of the options to define an event as an adverse event of special interest. However, the event 'stop of antirheumatic treatment for AE' is also taken into account as potential harm confounder in the analyses. We deleted this event from the definition of AE of special interest because we don't want to double count this event. So, the event "any AE (except loss of efficacy, worsening of disease) that leads to the definite cessation of one of the antirheumatic drugs, including trial medication" was changed to "any AE (except loss of efficacy, worsening of disease) that leads to the definite cessation of trial medication".
- 'Infection requiring antibiotic treatment' was discussed because the definition is not clear about topical treatments, and treatments for fungi and viruses. Therefore, we decided that:
  - For the purpose of classification, 'antibiotic' includes any specific treatment aimed at microorganisms to treat an infection: so this includes topical, antiviral, antifungal, antiparasitic treatment.
  - (Surgical) procedures with concomitant antibiotics: not (initially) an infection, so not AESI; AESI only when the procedure was done for a primary infection (e.g. abscess).
     Surgical complications treated with antibiotics are also not coded as AESI, because it is usually impossible to determine whether the antibiotic was given as prophylaxis or as treatment.

Note: any surgery is of necessity (hospital admission) already an SAE.

- A cardiovascular event (myocardial infarction, cerebrovascular event, peripheral arterial vascular event);
  - Anything falling outside this definition is not an AESI.
     So venous hemorrhoids, venous ulcus cruris, thrombosis, pulmonary embolism, subdural hematoma, and traumatic hemorrhagic brain lesions are not coded as AESI.
     Also cardiac rhythm disturbances, valve lesions, cardiac insufficiency, cardiomyopathy, and encephalopathy, are not coded as AESI unless part of an acute ischemic episode.
- Newly occurring hypertension requiring drug treatment;
- Newly occurring diabetes mellitus requiring drug treatment;
- Symptomatic bone fracture requiring treatment;
  - AESI is coded as 'no' if the vertebral fracture was asymptomatic, and 'yes' for all nonvertebral fractures, unless expressly indicated that the fracture was asymptomatic.
    - Note that vertebral fracture is also captured as secondary outcome through DEXA or spine radiographs.

- Newly occurring cataract or glaucoma.
  - Cataract and glaucoma are assumed to be bilateral.
     A medical history of the disease in one eye counts for both, so no AESI during the trial for procedures on the contralateral eye. We count bilateral procedures for new disease as one (not two) AESI.
- "Newly occurring diabetes or hypertension": no problems in adjudication.

# 10.2 Secondary endpoints

The measurements severity and duration of fatigue due to RA are included in the initial protocol, but not in the assessment. Severity of fatigue is part of the RA Impact of Disease (RAID) questionnaire and will be reported as described in section 1.4.2. Duration of fatigue was not included in the assessment and will not be reported.

The number of patients retained on study drug over time was not described as secondary endpoint in the protocol. However, this proportion is measured and will be presented with survival analysis.

# 12 Appendix C. Report of blinded data review meetings

Blinded Review of deviations leading to exclusion from the Per-Protocol Analysis

Report of Review Meetings 9 June, 14 July, 17 November 2020 and 8 February 2021. Final version dd 2 March 2021.

Attendees: Maarten Boers (PI/MM), Linda Hartman (PhD candidate), Hans Bijlsma (SAC member), Nick van der Bulk (CR2O, Head Clin Ops), Liza Bakker (sr. CRA), Linda Doerwald (Linical, Program Data manager), Leonie Middelink (Ops lead Gloria)

## **Documents used**

- Clinical study protocol version 4.0 12 February 2019
- Medical monitor plan dd. 05 April 2018
- PD tacker dd. 18 February 2021
- Manual listings 11 February 2021

## 1. Investigational Medicinal Product (IMP) deviations

The list of patients missing >20% of capsules per period (up to 3 months and up to 24 months) was reviewed. It was agreed that for the Per Protocol (PP) population adherence of at least 80% up to 3 months is required.

#### Review list:

- 1. Adherence should be at least 80% first 3 months done (between baseline and V2), if adherence is < 80%, the patients are excluded from the PP group. For the complete overview, see attachment PP vs ITT overview.
- 2. The periods of non-compliance after 3 months up to 24 months are left out of scope as they do not influence the PP population that applies only to the first 3 months.

#### 2. Protocol Deviations

The PD tracker (dd 04 Feb 2021, later updated with version 18 February 2021) was reviewed, and following deviations were discussed:

## Possible unblinding

Patients 107005 and -021 opened the capsules themselves.

As the unblinding took place in the first 3 months, they are out of the PP group.

Patient 107005 ICF signed on 31 Jan 2017, unblinding 24 Mar 2017; 107021 ICF signed on 22 aug 2018 and unblinding 6 Nov 2018

#### Prednisone open label use

The PD tracker was reconciled with the Conmeds page in the manual listings. This has been done after final coding. This list has been crossed checked with the PD tracker, and for all prohibited prednisolone open label use an PD form has been created. If this prohibited open label use took place in the 30 days before baseline, or between ICF signature date and V2, the patient is excluded

from the PP population (see prohibited meds sections). Other prednisolone open label use (after V2) will be flagged for analysis, but does not affect the PP selection.

In the coded conmeds file, the H02 ATC codes were selected. And the following rules were applied:

- IV GCs are always a Protocol Deviation (if before stop of IMP).
- Oral GCs are allowed for a maximum period of 3 weeks, for max 4 times, during IMP use.
- Intra-Articular and Intra Bursal are allowed a maximum of 4 times during IMP use
- Intra Muscular GCs are allowed to a maximum of 2 times during IMP use.

#### IMP deviations

If a patient misses a substantial percentage of the doses in a certain period (e.g. patient 116004 and 501009) after month 3, this does not affect the PP population, see above.

#### Time window deviations

As the time window deviations all have taken place after V2, this does not affect the PP evaluation.

#### Missed assessments

Only missing DAS-scores during the first 3 months of the trial will lead to exclusion from PP. A DAS28-CRP can be used instead of the DAS28ESR. It was decided not to impute the DAS-ESR with a RAPID3. For the following visits the DASESR will be imputed with a DASCRP.

| PatiëntID | Imputation | Visite |
|-----------|--------------------------------|--------|
| 104016 | DAS28ESR imputed with DAS28CRP | 2 |
| 106004 | DAS28ESR imputed with DAS28CRP | 2 |
| 110002 | DAS28ESR imputed with DAS28CRP | 1 |
| 110004 | DAS28ESR imputed with DAS28CRP | 2 |
| 113007 | DAS28ESR imputed with DAS28CRP | 2 |
| 113010 | DAS28ESR imputed with DAS28CRP | 1 |
| 114013 | DAS28ESR imputed with DAS28CRP | 2 |
| 117006 | DAS28ESR imputed with DAS28CRP | 2 |

## **Process deviations**

Deviations such as SAE timelines, ICF signatures etc. do not lead to exclusion.

## Eligibility criteria

All the deviations regarding eligibility criteria have been reviewed. Patients with actual deviations regarding violation of selection criteria are excluded from the PP. Process deviations relating to e.g. the Informed Consent process will not.

#### 3. Other RA medication

The type of medication, timing and exposure to the RA medication next to the IMP has been reviewed based on the manual listings.

The objective of the PP analysis in the first three months is to study the effects of low-dose prednisolone in a population without co-interventions. As the impact of concurrent RA med use is so substantial, patients who start or change prohibited meds (biologicals, DMARDs, GCs) between ICF and V2 of the trial are excluded from the PP population as well. As per protocol, start with other RA meds was not absolutely prohibited, we changed the term "per protocol population", "per protocol population, also excluding initial changes in antirheumatic medication". This terminology has also been updated in the final SAP.

#### 4. Other reviews to consider

- Safety reporting: cases of increase in disease activity (DA) were reported as AEs. No increase in DA reported as AE (based in coding file 5feb2021). Discussion pat 104008, AE# 9, swollen ancle left and right (NB site 114 3x painful joints / knee). All these AEs have been queried and the site confirmed it was an actual separate AE.
- The check of efficacy data for patients with an early end of treatment has been incorporated in the SAP.

The wording of the definitions of AEs of SI has been finetuned. Although this does not affect the PP evaluation, this has been discussed (as well as with the SAC), and the new rules for stop of RA meds and "anti-biotics" are to be applied after data export and before analysis. This has also been added to the SAP in the section "deviations from protocol".

The final list of patients included in the PP population is shown in Appendix D, below.

# 13 Appendix D. Gloria final PP population, also excluding initial changes in antirheumatic medication

| IMP <3 m | Possible unblinding | Prohib pred use | Missed<br>Ass | Eligibility<br>Vio | Other RA<br>meds ICF-V2 | Final |
|---|---|---|---|---|---|---|
| In | | | | Out | Out | Out |
| In | | | | | | |
| In | | | | Out | Out | Out |
| In | | | | | | |
| Out | | | DAS28 v2 | | Out | Out |
| In | | | DAS28 v2 | Out | | Out |
| In | | | | | | |
| In | | | DAS28 V2 | | | Out |
| In | | | | | | |
| In | | | | | | |
| Out | | | | | | Out |
| Out | | | DAS28 v2 | | Out | Out |
| In | | | | | Out | Out |
| In | | | | | | |
| In | | | | | | |
| In | | | | | | |
| In | | | DAS28 v1 | | Out | Out |
| Out | | | DAS28 v2 | Out | Out | Out |
| In | | | | | Out | Out |
| In | | | | | Out | Out |
| In | | | | | | |
| In | | | | | | |
| In | | | | | | |
| In | | | | | | |
| In | | | | | Out | Out |
| In | | | | | | |
| In | | | | | | |
| Out | | | | | | Out |
| In | | | | | | |
| In | | | | | Out | Out |
| In | | | | | | |
| In | | | | | | |
| In | | | | | | |
| In | | | | | | |
| In | | | | | | |
| | | | | | Out | Out |
| | | | | | Juc | Jul |
| | | | | | Out | 0 |
| | | | | | Out | Out |
| | In In In In Out In | In In In In In In In In | In | In | Unblinding Use Ass Vio Out | In |

| Patient | IMP <3 m | Possible unblinding | Prohib pred use | Missed<br>Ass | Eligibility<br>Vio | Other RA<br>meds ICF-V2 | Final |
|---|---|---|---|---|---|---|---|
| 102003 | In | | | | | | |
| 102004 | In | | | | Out | Out | Out |
| 102005 | Out | | | | | | Out |
| 102006 | In | | | | | | |
| 102007 | In | | | | | | |
| 102008 | In | | | | | | |
| 102009 | In | | | | | | |
| 104001 | In | | | | | Out | Out |
| 104004 | In | | | | | Out | Out |
| 104005 | In | | | | | | |
| 104006 | In | | | | | | |
| 104007 | In | | | | | Out | Out |
| 104008 | In | | | | | | |
| 104009 | In | | | | | | |
| 104010 | In | | | | | | |
| 104011 | In | | | | | Out | Out |
| 104012 | In | | | | | | |
| 104013 | In | | | | | | |
| 104014 | In | | | | | Out | Out |
| 104015 | In | | | | | Out | Out |
| 104016 | In | | | | | Out | Out |
| 104017 | In | | | | | | |
| 104018 | In | | | | | | |
| 104019 | In | | | | | | |
| 106001 | In | | | | | Out | Out |
| 106002 | In | | | | | | |
| 106003 | In | | | | | | |
| 106004 | In | | | | | | |
| 106005 | In | | | | | | |
| 106006 | In | | | | | | |
| 106007 | In | | | | | Out | Out |
| 106008 | In | | | | | | |
| 107001 | In | | | | | | |
| 107002 | In | | GC use first 3 months | | | Out | Out |
| 107003 | In | | | | | | |
| 107004 | In | | | | | | |
| 107005 | In | Unblinding < m3 | | DAS28 v2 | | | Out |
| 107006 | In | | | | | | |
| 107007 | Out | | | DAS28 v2 | | | Out |
| 107008 | In | | | | | | |
| 107009 | In | | | DAS28 v2 | | Out | Out |
| 107010 | In | | | | | | |
| 107011 | In | | | | | Out | Out |
| 107012 | In | | | | | | |
| 107013 | In | | | | | Out | Out |

| Patient | IMP <3 m | Possible unblinding | Prohib pred use | Missed<br>Ass | Eligibility<br>Vio | Other RA<br>meds ICF-V2 | Final |
|---|---|---|---|---|---|---|---|
| 107014 | In | | | | | Out | Out |
| 107015 | In | | | | | Out | Out |
| 107016 | In | | | | | | |
| 107018 | In | | | | | | |
| 107019 | In | | | | | Out | Out |
| 107020 | In | | | | | Out | Out |
| 107021 | In | Unblinding < m3 | | | | | Out |
| 107022 | In | | | | | | |
| 107023 | In | | | | | Out | Out |
| 107024 | In | | | | | Out | Out |
| 108001 | In | | | | | | |
| 108002 | In | | | | | | |
| 108003 | In | | | | | Out | Out |
| 108004 | In | | | | | | |
| 108005 | In | | | | | | |
| 108006 | Out | | | DAS28 v2 | | Out | Out |
| 108007 | In | | | | | | |
| 108008 | In | | | | | | |
| 108009 | In | | | | | | |
| 108010 | In | | | | | | |
| 108011 | In | | | | | | |
| 108012 | Out | | | | | | Out |
| 108013 | In | | | | | | |
| 108014 | In | | | | | | |
| 108015 | Out | | | DAS28 v2 | | | Out |
| 108016 | In | | | | | | |
| 108017 | In | | | | | | |
| 108018 | In | | | | | | |
| 108019 | Out | | | DAS28 v2 | | Out | Out |
| 108020 | Out | | | | | Out | Out |
| 108021 | In | | | | | Out | Out |
| 108022 | In | | | | | | |
| 108023 | In | | | | | Out | Out |
| 108024 | In | | | | | | |
| 108025 | Out | | | | | | Out |
| 108026 | In | | | | | Out | Out |
| 108027 | Out | | | DAS28 v2 | | Out | Out |
| 108027 | In | | | 5, 1320 VZ | | | Jul |
| 108029 | In | | | | | | |
| 108029 | In | | | | | | |
| 108030 | In | | | | | Out | Out |
| 108031 | In | | | | | Out | Out |
| 108032 | | | | DAS28 v2 | | Out | Out |
| | In | | | DA326 VZ | | | |
| 108034 | In | | | | | Out | Out |
| 108035 | Out | | | | | Out | Out |
| 108036 | In | | | | | | |

| Patient | IMP <3 m | Possible unblinding | Prohib pred use | Missed<br>Ass | Eligibility<br>Vio | Other RA meds ICF-V2 | Final |
|---|---|---|---|---|---|---|---|
| 108037 | In | | | | | | |
| 108038 | In | | | | | Out | Out |
| 108039 | Out | | | DAS28 v2 | | Out | Out |
| 108040 | In | | | | | Out | Out |
| 108041 | In | | | | | | |
| 108042 | Out | | | | | | Out |
| 108043 | In | | | | | Out | Out |
| 109001 | In | | | | | | |
| 109002 | In | | | | | Out | Out |
| 109003 | In | | | | | | |
| 109004 | In | | | | | | |
| 109005 | In | | | | | | |
| 109007 | In | | | | | Out | Out |
| 109008 | In | | | | | | |
| 109009 | In | | | | | | |
| 109010 | In | | | | | | |
| 109011 | In | | | | | | |
| 109012 | In | | | | | Out | Out |
| 109013 | In | | | | | Out | Out |
| 109014 | In | | | | | | |
| 109015 | In | | | | | Out | Out |
| 109016 | Out | | | | | | Out |
| 109017 | In | | | | | | |
| 109018 | In | | | | | | |
| 109019 | In | | | | | Out | Out |
| 110001 | In | | | | | | |
| 110002 | In | | | | | | |
| 110003 | In | | | | | | |
| 110004 | In | | | | | | |
| 110005 | In | | | | | | |
| 110006 | Out | | | DAS28 v2 | | | Out |
| 110007 | Out | | | | | | Out |
| 110008 | In | | | | | Out | Out |
| 110009 | In | | | | | | |
| 110010 | Out | | | | | | Out |
| 111001 | In | | | | | | |
| 111002 | In | | | | | | |
| 111003 | In | | | | | | |
| 111004 | In | | | | | | |
| 111005 | In | | | | | | |
| 111006 | In | | | | | | |
| 111007 | In | | | | | | |
| 111008 | In | | | | | | |
| 111009 | In | | | | | | |
| 112001 | In | | | | | | |
| 112002 | In | | | | | | |
| 112003 | In | | | | | | |

| Patient | IMP <3 m | Possible unblinding | Prohib pred use | Missed<br>Ass | Eligibility<br>Vio | Other RA meds ICF-V2 | Final |
|---|---|---|---|---|---|---|---|
| 112004 | In | | | | | | |
| 112005 | In | | | | | Out | Out |
| 112006 | In | | | DAS28 V2 | | | Out |
| 112007 | In | | | | | | |
| 112008 | Out | | | | | | Out |
| 112009 | In | | | | | | |
| 112010 | In | | | | | | |
| 112011 | In | | | | | | |
| 112012 | In | | | | | | |
| 112013 | In | | | | | | |
| 112014 | In | | | | | | |
| 112015 | In | | | | | Out | Out |
| 112016 | In | | | | | Out | Out |
| 112017 | In | | | | | | |
| 112018 | In | | | | | | |
| 112019 | In | | | | | Out | Out |
| 112020 | In | | | | | | |
| 112021 | In | | | | | Out | Out |
| 112022 | In | | | | | | |
| 112023 | In | | | | | | |
| 112024 | In | | | | | | |
| 112025 | In | | | | | | |
| 112026 | In | | | | | | |
| 112027 | In | | | | | | |
| 112028 | In | | | | | | |
| 112029 | In | | | | | | |
| 112030 | In | | | | | Out | Out |
| 112031 | In | | | | | | |
| 112032 | In | | | | | | |
| 112033 | In | | Pred < 30d<br>baseline | | | | Out |
| 112034 | In | | | | | | |
| 112035 | In | | | | | | |
| 112036 | In | | | | | | |
| 112037 | Out | | | | | | Out |
| 112038 | Out | | | | | | Out |
| 112039 | In | | Pred < 30d<br>baseline | | | Out | Out |
| 112040 | In | | | | | | |
| 112041 | In | | | | | | |
| 112042 | In | | | | | Out | Out |
| 112043 | Out | | | DAS28 v2 | | | Out |
| 112044 | In | | | | | | |
| 112045 | In | | | DAS28V2 | | | Out |
| 112046 | In | | | | | | |
| 112047 | In | | | | | | |
| 112048 | Out | | | | | | Out |
| 112049 | In | | | | | | |

| Patient | IMP <3 m | Possible unblinding | Prohib pred use | Missed<br>Ass | Eligibility<br>Vio | Other RA<br>meds ICF-V2 | Final |
|---|---|---|---|---|---|---|---|
| 112050 | In | | | | | Out | Out |
| 112051 | In | | | | | | |
| 112052 | In | | | | | | |
| 112053 | In | | | | | | |
| 112054 | In | | | | | Out | Out |
| 113001 | In | | | | | | |
| 113002 | Out | | | DAS28 v2 | | | Out |
| 113003 | In | | | | | | |
| 113004 | In | | | | | | |
| 113005 | In | | | | | Out | Out |
| 113006 | In | | | | | Out | Out |
| 113007 | In | | | | | | |
| 113008 | In | | | | | | |
| 113009 | In | | | | | | |
| 113010 | In | | | | | Out | Out |
| 113011 | In | | | | | | |
| 113012 | In | | | DAS28 v2 | | Out | Out |
| 114001 | In | | | DAS28 v1 | | Out | Out |
| 114002 | In | | | | | | |
| 114003 | In | | | | | | |
| 114004 | In | | | | | Out | Out |
| 114005 | Out | | | | | | Out |
| 114006 | Out | | | | | | Out |
| 114007 | In | | | | | | |
| 114008 | In | | | | | | |
| 114009 | In | | | | | | |
| 114010 | In | | | | | Out | Out |
| 114011 | In | | | | | | |
| 114012 | In | | | | | Out | Out |
| 114013 | In | | | | | | |
| 114015 | In | | | DAS28V2 | Out | | Out |
| 114016 | In | | | | | | |
| 115001 | In | | | | | | |
| 115002 | In . | | | | | | |
| 115003 | In . | | | | | | |
| 116001 | In . | | | | | | |
| 116002 | In . | | | | | | |
| 116003 | In . | | | | | | |
| 116004 | In . | | | | Out | | Out |
| 116005 | In . | | | | | | |
| 116006 | In . | | | | | | |
| 116007 | In . | | | | | | |
| 116008 | In . | | | | | | |
| 116009 | In . | | | | | | |
| 116010 | In | | | | | | |
| 116011 | Out | | | DAS28 v2 | | | Out |
| 116012 | In | | | | | | |

| Patient | IMP <3 m | Possible unblinding | Prohib pred<br>use | Missed<br>Ass | Eligibility<br>Vio | Other RA<br>meds ICF-V2 | Final |
|---|---|---|---|---|---|---|---|
| 116013 | In | | | DAS28 v2 | | | Out |
| 116014 | In | | | | | | |
| 116015 | In | | | | | | |
| 117001 | In | | | | | | |
| 117002 | In | | | | | | |
| 117003 | In | | | | | Out | Out |
| 117004 | In | | | | | | |
| 117005 | In | | | | | | |
| 117006 | In | | | | | | |
| 117007 | In | | | | | | |
| 117008 | In | | | | | | |
| 117009 | In | | | | | | |
| 117010 | In | | | | | | |
| 201001 | In | | | | | | |
| 201002 | In | | | | | | |
| 204001 | Out | | | DAS28 v2 | | | Out |
| 204002 | In | | | | | | |
| 204003 | In | | | | | | |
| 204004 | In | | | | | | |
| 204005 | In | | | | | | |
| 204006 | In | | | | | | |
| 204007 | In | | | | | | |
| 205001 | Out | | | | | Out | Out |
| 301001 | In | | | | | | |
| 301002 | In | | | | | | |
| 301003 | In | | | | | | |
| 301004 | In | | | | | | |
| 301005 | In | | | | | | |
| 301006 | Out | | | DAS28 v2 | | | Out |
| 301007 | In | | | | | | |
| 301008 | In | | | | | | |
| 301009 | In | | | DAS28 V2 | | | Out |
| 302001 | In | | | | | | |
| 303001 | In | | | | | | |
| 304001 | In | | | | | | |
| 304002 | Out | | | | | | Out |
| 304003 | In | | | | | | |
| 304004 | In | | | | | | |
| 304005 | In | | | | | | |
| 304006 | In | | | | | | |
| 304007 | Out | | | | | | Out |
| 304008 | In | | | | | | |
| 305001 | In | | | | | | |
| 305002 | In | | | | | | |
| 305003 | In | | | | | | |
| 305004 | In | | | | | | |
| 305005 | In | | | | | | |

| Patient | IMP <3 m | Possible unblinding | Prohib pred use | Missed<br>Ass | Eligibility<br>Vio | Other RA meds ICF-V2 | Final |
|---|---|---|---|---|---|---|---|
| 305006 | In | | | | | Out | Out |
| 305007 | In | | | | | | |
| 401001 | In | | | | | | |
| 401002 | In | | | | | | |
| 501001 | In | | | | | | |
| 501002 | In | | | | | | |
| 501003 | In | | | | | | |
| 501004 | In | | | | | | |
| 501005 | In | | | | | | |
| 501006 | In | | | | | | |
| 501007 | In | | | | | | |
| 501008 | In | | | | | | |
| 501009 | In | | | | | | |
| 501010 | In | | | | | | |
| 501011 | In | | | | | | |
| 501012 | In | | | | | | |
| 501013 | In | | | | | | |
| 501014 | In | | | | | | |
| 501015 | In | | | | | | |
| 501016 | In | | | | | | |
| 501017 | In | | | | | | |
| 501018 | In | | | | | | |
| 501019 | In | | | | | | |
| 501020 | In | | | | | | |
| 501021 | In | | | | | | |
| 501022 | In | | | | | | |
| 501023 | In | | | | | | |
| 501024 | In | | | | | Out | Out |
| 501025 | In | | | | | | |
| 501026 | In | | | | | | |
| 501027 | In | | | | | | |
| 501028 | In | | | | | Out | Out |
| 501029 | In | | | | | | |
| 501030 | In | | | | | Out | Out |
| 501031 | In | | | | | | |
| 501032 | In | | | | | | |
| 501033 | In | | | | | | |
| 501034 | In | | | | | | |
| 501035 | In | | | | | Out | Out |
| 501036 | In | | | | | | |
| 501037 | In | | | | | | |
| 501038 | In | | | | | | |
| 501039 | In | | | | | | |
| 501040 | In | | | | | | |
| 501041 | In | | | | | | |
| 501042 | In | | | | | | |
| 501043 | In | | | | | Out | Out |

| Patient | IMP <3 m | Possible unblinding | Prohib pred use | Missed<br>Ass | Eligibility<br>Vio | Other RA meds ICF-V2 | Final |
|---|---|---|---|---|---|---|---|
| 501044 | In | | | | | | |
| 501045 | In | | | | | | |
| 501046 | In | | | | | | |
| 501047 | In | | | | | | |
| 501048 | Out | | | DAS28 v2 | | | Out |
| 501049 | In | | | | | | |
| 501050 | In | | | | | | |
| 501051 | Out | | | | | Out | Out |
| 501052 | Out | | | DAS28 v2 | | | Out |
| 501053 | In | | | | | | |
| 501054 | In | | | | | | |
| 501055 | Out | | | | | | Out |
| 501056 | In | | | | | | |
| 501057 | In | | | | | | |
| 501058 | In | | | | | | |
| 501059 | In | | | | | | |
| 501060 | In | | | | | | |
| 601001 | Out | | | DAS28 v2 | | | Out |
| 601002 | Out | | | DAS28 v2 | | | Out |
| 601003 | In | | | | | | |
| 601004 | In | | | | | | |
| 601005 | Out | | | DAS28 v2 | | Out | Out |
| 601006 | In | | | | | | |
| 601007 | In | | | | | | |
| 601008 | In | | | | | | |
| 601009 | Out | | | DAS28 v2 | | | Out |
| 601010 | In | | | | | | |
| 601011 | Out | | | DAS28 v2 | | | Out |
| 601012 | In | | | | | | |
| 701001 | In | | | | | | |
| 701002 | In | | | | | | |
| 701003 | In | | | | | | |
| 701004 | In | | | | | | |
| 701005 | In | | | | | | |
| 701006 | Out | | | DAS28 v2 | | | Out |
| 701007 | In | | | | | | |
| 701008 | In | | | | | | |
| 701009 | In | | | | | | |
| 701010 | Out | | | | | | Out |
| 701011 | In | | | | | | |
| 701012 | In | | | | | Out | Out |
| 701013 | In | | | | | | |
| 701014 | In | | | | | | |
| 701015 | In | | | | | | |
| 701016 | In | | | | | | |
| 701017 | In | | | | | | |
| 701018 | In | | | | | | |

| Patient | IMP <3 m | Possible unblinding | Prohib pred use | Missed<br>Ass | Eligibility<br>Vio | Other RA meds ICF-V2 | Final |
|---|---|---|---|---|---|---|---|
| 701019 | Out | | | DAS28 v2 | | | Out |
| 701020 | In | | | | | | |
| 701021 | Out | | | | | | Out |
| 701022 | In | | | | | | |
| 701023 | Out | | | | | | Out |
| 701024 | Out | | | DAS28 v2 | | Out | Out |
| 701025 | In | | | | | | |
| 701026 | In | | | | | Out | Out |
| 701027 | In | | | | | | |
| 701028 | In | | | | | | |
| 701029 | In | | | | | | |
| 701030 | Out | | | DAS28 v2 | | | Out |
| 701031 | In | | | | | | |
| 701032 | In | | | | | | |
| 701033 | Out | | | DAS28 v2 | | | Out |
| 701034 | In | | | | | | |
| 701035 | In | | | | | Out | Out |
| 701036 | In | | | | | | |
| 701037 | In | | | | | | |
| 701038 | In | | | | | | |
| 701039 | Out | | | DAS28 v2 | | | Out |
| 701040 | In | | | | | | |
| 701041 | In | | | | | | |
| 701042 | In | | | | | | |
| 701043 | In | | | | | | |
| 701044 | Out | | | | | Out | Out |
| 701045 | In | | | | | Out | Out |
| 702001 | Out | | | | | | Out |
| 702002 | In | | | | | | |
| 702003 | Out | | | DAS28 v2 | | | Out |
| 702004 | Out | | | | | | Out |
| 702005 | In | | | | | | |
| 702006 | In | | | | | | |
| 702007 | Out | | | | | | Out |
| 702008 | In | | | | | | |
| 702009 | In | | | | | | |
| 702010 | Out | | | | | | Out |
| 702011 | Out | | | | | | Out |
| total | 60 | 2 | 3 | 42 | 7 | 90 | 147 |